Statistical Analysis Plan Version 3 J1P-MC-KFAJ

A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of LY3471851 (NKTR-358) in Adults with Systemic Lupus Erythematosus

NCT04433585

Approval Date: 31 January 2023

# 1. Statistical Analysis Plan: J1P-MC-KFAJ: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of LY3471851 (NKTR-358) in Adults with Systemic Lupus Erythematosus

#### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: this document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

#### LY3471851

Study J1P-MC-KFAJ is a randomized, double-blind, placebo-controlled, Phase 2 study of LY3471851 (NKTR-358), designed to investigate the efficacy and safety of LY3471851 in adult patients with Systemic Lupus Erythemotosus.

Eli Lilly and Company Indianapolis, Indiana USA 46285 Protocol J1P-MC-KFAJ Phase 2

**Document ID: VV-CLIN-074563** 

## 2. Table of Contents

| Sec | Section | |
|---|---|---|
| 1. | Statistical Analysis Plan: J1P-MC-KFAJ: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of LY3471851 (NKTR-358) in Adults with Systemic Lupus Erythematosus | 1 |
| 2. | Table of Contents | 2 |
| 3. | Revision History | 11 |
| 4. | Study Objectives | 14 |
| 4.1 | | |
| 4.2 | 2. Secondary Objectives | 14 |
| CC | | |
| 5. | Study Design | 16 |
| 5.1 | 1. Summary of Study Design | 16 |
| 5.2 | 2. Method of Assignment to Treatment | 17 |
| 6. | A Priori Statistical Methods | 18 |
| 6.1 | 1. Determination of Sample Size | 18 |
| 6.2 | | 18 |
| CC | | |
| 6.4 | | |
| 6.5 | | |
| | 6.5.1. Primary Estimand | |
| | 6.5.3. Supportive Estimand for Primary and Secondary Objectives | |
| CI | 0.5.5. Supportive Estimated for Filmary and Secondary Objectives | 23 |
| 6.6 | 6. Definition of Populations | 24 |
| 6.7 | • | |
| | 6.7.1. Demographics and Baseline Characteristics | |
| | 6.7.2. Historical Illness and Preexisting Conditions | |
| 6.8 | | |
| 6.9 | 1 1 | |
| | 6.9.1. Corticosteroids | |
| 6.1 | 10. Treatment Compliance | 30 |
| 6.1 | 11. Handling of Dropouts or Missing Data | 30 |

| 6.12. Multicenter Studies |
|--------------------------------------------------|
| 6.13. Multiple Comparisons/Multiplicity |
| 6.14. Primary Endpoint/Estimand Analyses |
| 6.15. Secondary Endpoints/Estimand Analyses |
| CCI |
| 6.19. Safety Analyses |
| 6.19.1. Extent of Exposure |
| 6.19.2. Adverse Events |
| 6.19.2.1. Adverse Events |
| 6.19.2.2. Serious Adverse Events |
| CCI |
| CCI |
| 6.19.4. Injection Site Reaction |
| 6.19.5. Clinical Laboratory Evaluation |
| 6.19.5.1. Abnormal Hepatic Tests 42 |
| 6.19.5.2. Hematologic Changes |
| 6.19.5.3. Lymphocyte Subset Cell Counts |
| 6.19.5.4. Lipids Effects |
| 6.19.5.5. Renal Function Effects |
| 6.19.5.6. Elevations in Creatine Phosphokinase |
| 6.19.5.7. Serum Immunoglobulin Concentrations |
| 6.19.6. Vital Signs and Other Physical Findings |
| 6.19.7. Additional Safety Sections |
| 6.19.7.1. Symptoms of Depression (QIDS-SR16) |
| 6.19.7.2. Columbia Suicide Severity Rating Scale |
| 6.20. Other Analyses |
| 6.20.1. Subgroup Analyses |
| CCI |
| 6.20.3. Annual Report Analyses 49 |
| 6.20.4. Clinical Trial Registry Analyses |
| 6.22. Data Monitoring Committee |
| 0.22. Data Wolfforing Confidence |

| J1P-MC-KFAJ Statistical Analysis Plan Version 3 | | |
|-------------------------------------------------|-----------------|----|
| 7. | Unblinding Plan | 52 |
| 8. | References | 53 |
| 9. | Appendices | 54 |

| Table | of ( | Co | nte | nts |
|-------|------|----|-----|-----|
|-------|------|----|-----|-----|

| Table KFAJ.5.1. | Countries and Their Geographical Regions | 17 |
|---|---|---|
| Table KFAJ.6.1. | Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure<br>and Pulse Measurement, and Categorical Criteria for Weight Changes | |
| | for Adults. | 47 |

#### **Table of Contents**

| Figure | | Page |
|---|---|---|
| Figure 5.1. | Schema of Study J1P-MC-KFAJ, a Phase 2 study to evaluate the efficacy and safety of LY3471851 in adults with systemic lupus | |
| | erythematosus. | 16 |

#### **Table of Contents**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Description and Derivation of Efficacy Outcomes Measures and Endpoints | 55 |
| Appendix 2. | Description of Efficacy Analyses | 66 |
| Appendix 3. | Corticosteroid | 79 |
| Appendix 4. | List of MedDRA Preferred Terms for Potential Opportunistic Infections (POI) | 81 |
| Appendix 5. | List of MedDRA Preferred Terms for Elevated or Increased Lipids from the Dyslipidemia SMQ (SMQ 20000026) | 95 |
| Appendix 6. | List of Planned Laboratory Analytes with Reference Range Sources | 97 |
| Appendix 7. | Common Terminology Criteria for Adverse Events (CTCAE) Related to Myelosuppressive Events | 100 |

# **List of Abbreviations and Definitions of Terms**

| Term | Definition |
|----------|---------------------------------------------------------------|
| CCI | |
| AE | adverse events |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| Anti-HBc | hepatitis B core antibody |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BICLA | BILAG-based Composite Lupus Assessment |
| BILAG | British Isles Lupus Assessment Group – 2004 |
| CI | |
| CD | cluster of differentiation |
| CI | confidence interval |
| CLASI | Cutaneous Lupus Erythematosus Disease Area and Severity Index |
| CSR | clinical study report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTR | Clinical Trial Registry |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eDISH | evaluation of Drug-Induced Serious Hepatotoxicity |
| ETV | early termination visit |
| HbsAb | hepatitis B surface antigen |
| HbcAb | hepatitis B core antibody |
| HBV | hepatitis B virus |

| Term | Definition |
|--------|----------------------------------------------|
| HDL | high-density lipoprotein |
| IAC | internal assessment committee |
| ICE | intercurrent event |
| ICH | International Conference on Harmonisation |
| lg | immunoglobulin |
| IL | interleukin |
| IR | incidence rate |
| ISR | injection site reaction |
| IWRS | interactive web-response system |
| LCTPB | Large Clinical Trial Population Based |
| LDL | low-density lipoprotein |
| LLDAS | Lupus Low Disease Activity State |
| LS | least squares |
| LTT | Lowest Level Term |
| CCI | |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | modified intent-to-treat |
| MMRM | mixed models for repeated measures |
| NRI | nonresponder imputation |
| CCI | |
| NK | natural killer |
| NMSC | nonmelanoma skin cancers |
| CCI | |
| PEG | polyethylene glycolated |
| РК | pharmacokinetic |
| POI | potential opportunistic infections |

| Term | Definition |
|-----------|----------------------------------------------------------|
| PRO | patient-reported outcomes |
| PT | Preferred Term |
| PY | patient-year |
| Q2W | every 2 weeks |
| QIDS-SR16 | Quick Inventory of Depressive Symptomatology Self-Rated |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SLE | systemic lupus erythematosus |
| SLEDAI-2K | Systemic Lupus Erythematosus Disease Activity Index 2000 |
| SLEDAI-4 | a ≥4-point reduction in SLEDAI-2K score from baseline |
| SMQ | Standardised MedDRA Query |
| soc | System Organ Class |
| SRI-4 | Systemic Lupus Erythematosus Responder Index-4 |
| CCI | |
| TEAE | treatment-emergent adverse events |
| ULN | upper limit of normal |







# 4. Study Objectives

## 4.1. Primary Objective

| Objectives | Endpoints/Estimands |
|---|---|
| To determine whether treatment with LY3471851<br>Q2W is superior to placebo in reducing the signs<br>and symptoms of SLE as measured by SLEDAI-4 | • The study will compare LY3471851 with placebo in participants with SLE. |
| | <ul> <li>The primary comparison of interest is the difference<br/>in proportion of participants who achieve<br/>SLEDAI-4 response at Week 24.</li> </ul> |
| | The primary comparison will be assessed using a composite estimand where the intercurrent events of premature discontinuation and use of prohibited medication are part of the response definition. |

Abbreviations: Q2W = every 2 weeks; SLE = systemic lupus erythematosus; SLEDAI-4 = a ≥4-point reduction in SLEDAI-2K score from baseline; SLEDAI-2K = Systemic Lupus Erythematosus Disease Activity Index 2000.

## 4.2. Secondary Objectives

The secondary objectives of the study are the following:

| Objectives | Endpoints/Estimands |
|---|---|
| To determine whether treatment with LY3471851 Q2W is superior to placebo in reducing other measures of signs and symptoms of SLE | The study will compare LY3471851 with placebo in participants with SLE. |
| | Secondary comparisons of interest are the difference in proportion of participants who at Week 24 (V15) achieve: BILAG-based Composite Lupus Assessment (BICLA) response SRI-4 response |
| | <ul> <li>Lupus Low Disease Activity State (LLDAS)</li> <li>Secondary objectives will be assessed using a composite estimand.</li> </ul> |
| To characterize the pharmacokinetics of<br>LY3471851 in participants with SLE | LY3471851 plasma trough concentrations at Week 24 (V15) |

Abbreviations: BILAG = British Isles Lupus Assessment Group – 2004; Q2W = every 2 weeks; SLE = systemic lupus erythematosus; SRI-4 = Systemic Lupus Erythematosus Responder Index-4; V = Visit.



## 5. Study Design

#### 5.1. Summary of Study Design

Study KFAJ is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 2 study to evaluate the efficacy and safety of LY3471851 in adult study participants with at least moderately active SLE. The study has 3 required study periods and an optional prescreening period. A schematic of the study design is presented in Figure 5.1.



Note: Visit 802 is for HBV DNA testing of randomized participants who were positive for antibody to hepatitis B core antigen (anti-HBc) at screening.

Abbreviations: anti-HBc = hepatitis B core antibody; FD = first dose administered; HBV = hepatitis B virus; LD = last dose administered; Q2W = every 2 weeks; V = eCRF visit; W = study week relative to baseline visit.

Figure 5.1. Schema of Study J1P-MC-KFAJ, a Phase 2 study to evaluate the efficacy and safety of LY3471851 in adults with systemic lupus erythematosus.

**Optional prescreening period:** The optional prescreening period is prior to Visit 1. The optional prescreening visit (Visit 601) is intended for those investigators who opt for central laboratory assessment of the prospective participant's antinuclear antibodies, anti-double stranded DNA, and anti-Smith antibody status before full screening activities are initiated. The prescreening visit can be repeated 2 times (no more) per participant, with a minimum of 4 weeks between visits.

**Screening period:** The required screening period begins with Visit 1, which occurs within 5 weeks before the planned randomization visit (Week 0, Visit 2). Participants found to be eligible according to all of the study entry criteria will be randomly assigned in a 1:1:1:1 ratio to receive one of the following study interventions:

- CCI LY3471851 Q2W
   CCI LY3471851 Q2W
   CCI LY3471851 Q2W, and
- placebo Q2W.

Participants will be stratified at randomization according to disease activity at baseline, corticosteroid dose at baseline, and geographic region (Section 5.2). Study interventions will be administered via subcutaneous injection.

**Double-blind treatment period:** Randomized participants will begin the double-blind, placebo-controlled, 24-week treatment period at Visit 2. Participants will receive the first dose of the assigned study intervention at that visit and will continue to receive doses through the last scheduled dosing visit specified in protocol. Participants will maintain their usual standard-of-care medication regimen for SLE and for other diseases throughout the study, unless these medication regimens are specifically excluded by the study entry criteria. Safety and efficacy assessments and laboratory sample collections will be performed as specified in the protocol.

**Follow-up period:** All participants will have a posttreatment follow-up visit (Visit 801) for safety assessments. Randomized participants who were positive for anti-HBc at screening will have one additional posttreatment follow-up visit (Visit 802).

**Early discontinuation:** Participants who permanently discontinue the study drug early or withdraw from the study will undergo early termination procedures, including an ETV and the post-treatment follow-up visits specified in the protocol.

#### 5.2. Method of Assignment to Treatment

Subjects who meet all criteria for enrollment will be randomized 1:1:1:1 to double-blind treatment at Visit 2. Participants will be stratified at randomization according to disease activity at baseline (SLEDAI-2K <10; SLEDAI-2K ≥10), corticosteroid dose at baseline (<10 mg/day or ≥10 mg/day), and geographic region. Table KFAJ.5.1 describes how each region will be defined for the stratification at randomization as well as the statistical analyses and summaries.

Assignment to treatment groups will be determined by a computer-generated random sequence using an IWRS. The IWRS will be used to assign vials containing double-blind investigational product to each patient. Site personnel will confirm that they have located the correct vials by entering a confirmation number found on the vials into the IWRS. The IWRS will be used to assign investigational product to each patient. Site personnel will confirm that they have located the correct packages by entering a confirmation number found on packages into the IWRS.

 Table KFAJ.5.1.
 Countries and Their Geographical Regions

| Geographical Region | Country or Countries |
|---|---|
| North America | Canada, United States, Puerto Rico |
| Latin America | Argentina, Mexico |
| Europe | Belgium, Czech Republic, France, Germany, Hungary, Italy, Poland, Romania, Spain, United Kingdom |
| Asia | South Korea, Taiwan |
| Japan | Japan |
| Rest of World | Australia, India, Israel, Russia, Ukraine |

#### 6. A Priori Statistical Methods

#### 6.1. Determination of Sample Size

will be randomly assigned to study intervention. All randomized participants in the mITT population as defined in Section 6.6 will be considered evaluable.

Pairwise 2-sided tests of proportions with alpha = 0.05 will be performed on each LY3471851 dose versus placebo cell and a placebo response of 0.40, and a LY3471851 response of 0.64 for the maximally efficacious LY3471851 dose, there is at least 80% power to detect a statistically-significant difference in SLEDAI-4 response between LY3471851 and placebo at Week 24 (Visit 15).

#### 6.2. General Considerations

Statistical analysis of this study will be the responsibility of the sponsor or its designee. For primary and key secondary objectives, statistical analyses will be performed CCI

Not all displays described in this SAP will necessarily be included in the CSR. Not all displays will necessarily be created as a "static" display. Some may be incorporated into interactive display tools such as Spotfire instead of, or in addition to, a static display. Any display described in this SAP and not included in the CSR would be available upon request.

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, unless otherwise stated. The p-values will be rounded up to 3 decimal places. For example, any p-value strictly >0.049 and  $\le 0.05$  will be displayed as 0.050. This guarantees that on any printed statistical output, the unrounded p-value will always be less than or equal to the displayed p-value. A displayed p-value of 0.001 will always be understood to mean  $\le 0.001$ . Likewise, any p-value displayed as 1.000 will be understood to mean >0.999 and  $\le 1$ .

The primary analysis method for treatment comparisons of categorical efficacy and health outcome variables will be made using a logistic regression analysis with treatment group, baseline disease activity (SLEDAI-2K <10; SLEDAI-2K ≥10), corticosteroid dose at baseline (<10 mg/day or ≥10 mg/day), and geographic region (North America, Latin America, Europe, Asia, Japan, Rest of World) in the model. For each treatment comparison, an estimate of the treatment difference with corresponding Wald 95% CI, the odds ratio with corresponding Wald 95% CI and p-value will be presented. Each treatment group will be compared to the placebo group. The p-value for all other explanatory variables will also be presented. When logistic regression sample size requirements are not met (<5 subjects in any category for any factor), treatment comparison will be performed using the Fisher's exact test.

The primary analyses for continuous efficacy and health outcome variables will be made using MMRM. When MMRM is used, the model will include treatment, baseline score, baseline disease activity (SLEDAI-2K <10; SLEDAI-2K ≥10), corticosteroid dose at baseline (<10 mg/day or ≥10 mg/day), geographic region (North America, Latin America, Europe, Asia, Japan, Rest of World), visit (as categorical variable), the interaction of treatment-by-visit, and

the interaction of baseline value-by-visit as fixed factors. An unstructured covariance matrix will be used to model the within-patient variance-covariance errors. If this analysis fails to converge, the following structures will be tested in this pre-specified order: 1) heterogeneous Toeplitz, 2) heterogeneous autoregressive, 3) heterogeneous compound symmetry, 4) Toeplitz, 5) autoregressive), and 6) compound symmetry. The first covariance structure that converges using this prespecified order will be used. The Kenward-Roger method will be used to estimate the degrees of freedom. Type III sums of squares for the LS means will be used for the statistical comparison. The LS mean for each treatment group along with the estimate of the difference between treatments (difference between each LY3471851 dose group and placebo), standard error, p-value, and the 95% CIs will be reported at each visit along with p-values. For variables that are not collected at each postbaseline visit, data may exist at visits where the variable was not scheduled to be collected, due to early discontinuation visits. In these situations, data from the early discontinuation visit that do not correspond to the planned collection schedule will be excluded from the MMRM analyses (Andersen and Millen 2013). However, the data will still be used in other analyses.

When ANCOVA is used for efficacy/Health Outcomes measures, the model will include treatment, baseline score, baseline disease activity (SLEDAI-2K <10; SLEDAI-2K ≥10), corticosteroid dose at baseline (<10 mg/day or ≥10 mg/day), and geographic region as fixed factors. Type III sums of squares will be used. Differences in LS means between treatment groups will be displayed, with the p-value associated with the LS mean comparison to placebo (for each LY3471851 dose group) along with the 95% CI of the LS mean difference also provided. In addition to the LS means and tests, mean, SD, minimum, first quartile, median, third quartile, and maximum will be displayed.

When Cox regression is used for time-to-event variables, the model will include treatment, baseline score, baseline disease activity (SLEDAI-2K <10; SLEDAI-2K  $\ge$ 10), corticosteroid dose at baseline (<10 mg/day or  $\ge$ 10 mg/day) and geographic region (North America, Latin America, Europe, Asia, Japan, Rest of World). Treatment comparisons will use the hazard ratios and corresponding p-values from the Cox regression. The Kaplan-Meier product limit method will be used to estimate the survival curves for time-to-event variables. Patients completing the treatment period without event will be censored at the date of completion. Patient without an event, a date of completion, or discontinuation for the treatment period will be censored at the latest nonmissing date out of the following dates: date of last dose and date of last attended visit in the treatment period. Under the hypothetical estimand strategy, patients without an event prior to the first violation of concomitant medication rules will be censored at the time of the first violation of concomitant medication rules.



Efficacy and PRO analysis models may contain the independent variables such as treatment group, baseline disease activity, and geographic region.

Any change to the data analysis methods described in the SAP will require an amendment only if the change affects a principal feature of the SAP. Any other change to the data analysis methods described in the SAP, and the justification for making the change, will be described in the CSR. Additional exploratory analyses of the data will be conducted as deemed appropriate.







#### 6.4. Definition of Baseline and Postbaseline Measures

Baseline will be defined as the last available value before the first dose of study drug for both efficacy and safety analyses, unless otherwise specified. In most cases, this will be the measure recorded at Week 0 (Visit 2). The treatment period starts after the first study drug administration and ends on one of the following:

- date of Visit 15 (Week 24) for patients who completed the treatment period
- for patients who discontinued treatment early
  - o date of ETV, if ETV occurs less than 42 days after treatment discontinuation
  - o date of the last visit that occurs less than 42 days after treatment discontinuation, if ETV occurs after 42 days since treatment discontinuation.

Change from baseline will be calculated as the visit value of interest minus the baseline value. Percent change from baseline will be calculated as 100 times change from baseline divided by baseline.

Postbaseline measurements are collected after study drug administration through Visit 15 (Week 24) or an early discontinuation visit. For electronic PROs related to efficacy assessments, unscheduled postbaseline visits that fall within the protocol-defined visit windows will be summarized in the by-visit analyses if there is no scheduled visit available. If more than 1 value is reported for the same scheduled visit, then the first value will be summarized in the by-visit analyses.

The Follow-up Period includes all visits that are 42 days or more after treatment discontinuation for patients who discontinue the treatment period early. For patients who complete the treatment period, the Follow-up Period includes Visit 801 for safety assessment. Randomized participants who were positive for anti-HBc at screening will have one additional posttreatment follow-up visit (Visit 802). The baseline value for the safety analysis of the posttreatment follow-up period is defined as the last nonmissing assessment prior to entering the posttreatment Follow-up Period, that is Week 24 (Visit 15) for treatment completers or last visit that occurred less than 42 days after treatment discontinuation for patients that discontinued treatment early. When the

Follow-up Period includes more than 1 visit, any safety analyses that are done for this period will only include the first visit of this period.

#### 6.5. Primary, Secondary, and Supportive Estimands

Unless otherwise specified, a composite strategy will be used for categorical efficacy endpoints, as described in Section 6.5.1. A hypothetical strategy will be used for continuous efficacy endpoints, as described in Section 6.5.4.

#### 6.5.1. Primary Estimand

The primary clinical question of interest is: What is the difference between LY3471851 and placebo in the target patient population, in achieving a successful response at Week 24 without violating concomitant medication rules?

The violation of concomitant medication rules for this study includes (i) initiating or increasing in dose of corticosteroids, antimalarial, or immunosuppressant, or (ii) using prednisone >10 mg per day (or equivalent) after Week 12.

The estimand for the primary objective is described by the following attributes:

- population: modified intent-to-treat population
- endpoint: SLEDAI-4 at Week 24
- how to account for ICEs: A <u>composite estimand strategy</u> will be used. Participants with violation of concomitant medication rules will be considered as treatment failure, that is, a nonresponder, after the first occurrence of violation of concomitant medication rules.
- population-level summary: difference in response rate of SLEDAI-4 at Week 24 between LY3471851 and placebo, and
- rationale for estimand: the primary estimand strategy assumes that a participant, who violates concomitant medications, was not receiving sufficient benefits from study intervention. This estimand is free of confounding effects of increase in concomitant medication use. Under the primary estimand strategy, a participant is considered a SLEDAI-4 responder at Week 24 if both of the following are met:
  - ≥4 points reduction from baseline in SLEDAI-2K score at Week 24
  - o no violation of concomitant medication rules prior to Week 24.

If either or both of these criteria are not met, a participant is considered as a SLEDAI-4 nonresponder at Week 24. Apart from the primary estimand strategy, missing data imputation is described separately in Section 6.11.

## 6.5.2. Secondary Estimands

The secondary estimands for the secondary objectives are described by the following attributes:

- population: mITT population
- endpoints: SRI-4 at Week 24, BICLA at Week 24 (in the subset of participants with ≥1 A or ≥2 B at baseline), LLDAS at Week 24

- ICE will be accounted using the same estimand strategy as for the primary estimand (Section 6.5.1).
- population-level summary: difference in response rate of a secondary endpoint between LY3471851 and placebo
- rationale for estimand is provided in Section 6.5.1.

#### 6.5.3. Supportive Estimand for Primary and Secondary Objectives

A supportive estimand for the primary and secondary objectives will be considered to address a clinical question: What is the difference between LY3471851 and placebo in the target patient population, in achieving successful response at Week 24 without regards to violation of concomitant medication rules?

For the supportive estimands, a <u>treatment policy estimand strategy</u> will be used to account for ICEs, and treatment effect will be assessed regardless of whether ICEs has occurred or not. That is, observed data after ICEs will be included as is in the analysis. Population, endpoints, and population-level summary are the same as described in Sections 6.5.1 and 6.5.2.





#### 6.6. Definition of Populations

The following populations are defined for this study:

| Population | Description |
|---|---|
| Entered population | All participants who sign the informed consent form |
| Modified Intent-to-Treat (mITT) population | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants will be analyzed according to the intervention to which they were assigned. |
| Per-Protocol (PP) population | All randomized patients who do not commit an Important Protocol Deviation (IPD) that could potentially compromise efficacy results. IPDs are specified in the Trial Issue Management Plan. |
| Safety population | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention and did not discontinue the study for the reason "lost to follow-up" at the first postbaseline visit. Participants will be analyzed according to the intervention they actually received within each study period. |
| Pharmacokinetic (PK) Analysis population | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention they actually received and have PK data available. |

The mITT population will be used in analyses of efficacy and PRO, unless otherwise specified.

## 6.7. Participant Characteristics

## 6.7.1. Demographics and Baseline Characteristics

Demographics and baseline characteristics will be summarized using the mITT population by treatment group. The summary will include descriptive statistics such as the number of patients (n), mean, SD, median, min, and max for continuous measures, and frequency counts and percentages for categorical measures. No formal statistical comparisons will be made among treatment groups, unless otherwise stated.

The continuous demographic and baseline characteristic variables outlined in Table KFAJ.6.1 will be summarized using descriptive statistics.

Table KFAJ.6.1. Continuous Demographic and Baseline Characteristic Variables

| Variable | Quantitative | Categorical Summary | Subgroup Analysis |
|---|---|---|---|
| Demographic Characteristic | es | | |
| Age a | Yes | <65, 65 to <75, ≥75 | |
| | | ,, | |
| Height | Yes | | |
| Weight | Yes | | |
| BMI b | Yes | | |
| Sex | No | Female, Male | Yes |
| Race | No | American Indian/Alaska Native, Asian,<br>Black/African American, Native<br>Hawaiian or other Pacific Islander,<br>White, or Multiple | Yes |
| Country | | Canada, United States, Puerto Rico,<br>Argentina, Mexico, Belgium, Czech<br>Republic, France, Germany, Hungary,<br>Italy, Poland, Romania, Spain, United<br>Kingdom, South Korea, Taiwan, Japan,<br>Australia, India, Israel, Russia, Ukraine | |
| Region (Table KFAJ.5.1) | | North America, Latin America,<br>Europe, Asia, Japan, Rest of World | Yes |
| Country GDP | No | Category 1 [Mexico, India, Ukraine] Category 2 [Argentina, Czech Republic, Hungary, Poland, Romania, Spain, Russia] Category 3 [Canada, United States, Puerto Rico, Belgium, France, Germany, Italy, United Kingdom, South Korea, Taiwan, Japan, Australia, Israel] | Yes |
| Ethnicity (only US sites) | | Hispanic/Latino, Non-Hispanic/Non-<br>Latino, Missing | Yes |
| Time since onset of lupus (years) <sup>c</sup> | Yes | | |
| Concomitant Medication Use | at Baseline | | <u>I</u> |
| Daily dose of prednisone (or equivalent) in mg/day d | Yes | <7.5 mg/day, ≥7.5 mg/day<br><10 mg/day, ≥10 mg/day | Yes |
| Immunosuppressant use | No | Yes, No | |
| Mycophenolate mofetil use | No | | |
| Azathioprine use | No | | |
| Methotrexate use | No | | |

| Variable | Quantitative | Categorical Summary | Subgroup Analysis |
|---|---|---|---|
| Antimalarial use (for each | No | Yes, No | |
| drug) | | | |
| NSAID use | No | | |
| Disease Severity at Baseline | | | |
| SLEDAI-2K | Yes | <10,≥10 | Yes |
| SLEDAI-2K organ system involvement at baseline | No | Yes, No | |
| British Isles Lupus Assessment Group (BILAG) organ system involvement at baseline (either A or B) | No | Yes, No | |
| BILAG A organ system involvement at baseline | No | Yes, No | Yes |
| CCI | | | |
| CCI | | | |
| CCI | | | |
| CCI | | | |
| CCI | Yes | | |
| Physician's Global Assessment of Disease Activity score | Yes | | |
| CCI | | | |
| CCI | | | |
| CCI | | | |

| Variable | Quantitative | Categorical Summary | Subgroup Analysis |
|---|---|---|---|
| SLE Risk Probability Index | Yes | $\leq$ 7, 7 to $\leq$ 11, 11 to $\leq$ 14, >14 (lower | Yes |
| (SLEPRI) | | bounds are strictly greater than) | |
| Prior Benlysta (belimumab) | No | Yes, No | |
| use | | | |



Abbreviations: GCI ; GDP = gross domestic product; NRS = numeric rating scale; NSAID = nonsteroidal anti-inflammatory drug; SLE = Systemic Lupus Erythematosus; SLEDAI-2K = Systemic Lupus Erythematosus Disease Activity Index 2000.

- a Age will be calculated using an imputed date of birth of July 1st in the year of birth collected in the electronic case report form (eCRF). It will be calculated as: Age (in years) = (date of first dose imputed date of birth)/365.25
- b Body mass index (BMI) (kg/m2) at Visit 2. BMI (kg/m<sup>2</sup>) = Weight [kg] / Height [m]<sup>2</sup>
- c Time since onset of lupus will be calculated using the date of onset of lupus (as recorded on the SLE History eCRF page) as follows: Time since onset of lupus (years) = (date of first dose date of onset of lupus + 1) / 365.25.



d Patients with a non-zero dose at Visit 2 will be included in this baseline summary, see Section 6.9.1 for details of prednisone (or equivalent) baseline dose.

## 6.7.2. Historical Illness and Preexisting Conditions

Historical illness/condition is defined as the condition/event recorded on the Pre-Existing Conditions and Medical History eCRF page or on the Prespecified Medical History eCRF page with an end date prior to the date of informed consent. Preexisting condition is defined as the condition/event recorded on the Pre-Existing Conditions and Medical History eCRF page or on the Prespecified Medical History eCRF page with a start date prior to the date of informed consent, and no end date (that is, the event is ongoing) or an end date on or after the date of informed consent. Notice if a preexisting condition worsens in severity on or after the date of informed consent, it will be recorded as an AE on Adverse Events eCRF page from the date of worsening onwards. Historical illnesses and preexisting conditions will be classified using the latest version of the MedDRA. The number and percentage of patients with historical illnesses and preexisting conditions will be provided by treatment group, overall and by SOC and PT using the mITT population. Note that conditions with a partial or missing start date will be assumed to be "not preexisting" unless there is evidence, through comparison of partial dates, to suggest otherwise. Patients will only be counted once if same PT is listed in 2 or more different SOC categories.

### 6.8. Participant Disposition

A detailed description of participant disposition will be provided, including a summary of the number and percentage of participants entered into the study and randomized, the number and percentage of participants who complete the study or discontinue, both overall and by reason for discontinuation, and the frequency and percentage of patients who discontinue study treatment. A summary of important protocol deviations will be provided.

## 6.9. Concomitant Therapy

Previous and concomitant medications will be summarized by treatment group and will be presented by ATC drug classes using the latest version of the World Health Organization drug dictionary.

Under the composite estimand strategy described in Section 6.5.1, a patient will be considered a nonresponder after the first occurrence of a violation of any of the following concomitant medication rules, regardless of the patient's efficacy status or disposition status:

- no initiation or increase in dose from baseline of
  - nonsteroidal anti-inflammatory drug intended for treatment of signs and symptoms of SLE
  - o prednisone (or equivalent)
  - o antimalarial, and
  - o immunosuppressant
- prednisone ≤10 mg/day (or equivalent) by Week 12

Violations of concomitant medication rules will be first identified via programming and then reviewed by a blinded medical to confirm the violations align with the criteria specified in the protocol. The confirmed list provided by the blinded medical will be used for analyses.

#### 6.9.1. Corticosteroids

To allow for assessments of changes in doses of various corticosteroids, it was necessary to standardize all corticosteroid doses to an equivalent prednisone dose. Table KFAJ.6.2 provides a summary of frequent corticosteroids and their prednisone-equivalent dose. The dose of the drug listed in Column 1 is multiplied by the conversion factor in Column 2 to provide the prednisone equivalent dose (in milligrams). This dose of corticosteroid will be referred to as "prednisone (or equivalent)" throughout this document.



See Appendix 3 for a complete table showing conversion factors for each corticosteroid medication identified during the study, instructions for selecting corticosteroids, and the manual review process. References for this table can also be found in Appendix 3.

Baseline prednisone (or equivalent) dose will be the total daily dose of all corticosteroids being taken by a patient at Visit 2. This baseline dose will be used for baseline summaries and for comparisons to later visits. A daily dose of prednisone (or equivalent) will be calculated for each day between baseline and treatment discontinuation. The daily dose of prednisone (or equivalent) at each visit date will be used as the corticosteroid dose for that visit.

#### 6.10. Treatment Compliance

Patient compliance with study medication will be assessed from the randomization visit (Week 0) to Visit 15 (Week 24) during the treatment period. Compliance will be summarized from randomization until end of treatment using the mITT population. A patient is considered noncompliant if 2 or more of the prescribed doses during the study are missed, not including doses withheld by the investigator. A patient who takes more than 12 of the prescribed doses during the treatment period is also considered noncompliant.

Compliance to study drug in the period of interest will be calculated as follows:

$$\frac{\text{actual total # of doses}}{\text{Expected total # of doses}} * 100.$$

If a patient has a dose temporarily interrupted by the investigator during the period, the total number of days that drug was withheld will be deducted from the total number of days in the calculation of the expected total number of doses used.

The summary statistics of the percent of compliance and noncompliance rate will be summarized by treatment group. The percent of compliance for Week 0 (Visit 2) through Week 24 (Visit 15) will be presented, along with the associated noncompliance rates.

### 6.11. Handling of Dropouts or Missing Data

Missing data imputation is handled separately from the estimand strategy. After intercurrent events are accounted for according to an estimand strategy described in Section 6.5, any remaining missing data will be handled using missing data imputation methods described in this section. Reasons for such missing data include, but are not limited to,

- intermittent missing visits, assessments, or some components of assessments
- temporary treatment interruptions, and
- early treatment discontinuation.

When NRI is used, missing binary data will be imputed as non-response.

When last observation carried forward is used, missing continuous data will be imputed with the last nonmissing postbaseline observation prior to the first occurrence of intercurrent events. For patients without at least one postbaseline observation, missing continuous data will not be imputed.

When baseline observation carried forward is used, missing continuous data will be imputed with baseline observation (last nonmissing data before the first injection). For patients without baseline observation, missing continuous data at postbaseline visits will not be imputed.

The missing data imputation methods for planned analyses are specified in Sections 6.14, 6.15, and 6.16.

#### 6.12. Multicenter Studies

This study will be conducted by multiple investigators at multiple sites internationally. The countries will be categorized into geographic regions, as described in Section 5.2. Geographic region will be included in a statistical model as a fixed effect, unless otherwise specified.

#### 6.13. Multiple Comparisons/Multiplicity

No adjustments for multiplicity will be made for any analyses in this study.

### 6.14. Primary Endpoint/Estimand Analyses

The primary efficacy endpoint per composite estimand strategy (the primary estimand as described in Section 6.5.1) is

• SLEDAI-4 at Week 24 after accounting for violation of concomitant medication rules: (i) initiating or increasing in dose of corticosteroids, antimalarial, or immunosuppressant, or (ii) using prednisone >10 mg per day (or equivalent) after Week 12

Under the composite estimand strategy, participants will be considered nonresponders at all subsequent visits after the first violation of concomitant medication rules regardless of their discontinuation status.

The primary analysis for treatment comparison of each LY3471851 dose with placebo will be analyzed using a logistic regression model with treatment group, baseline disease activity (SLEDAI-2K <10; SLEDAI-2K ≥10), corticosteroid dose at baseline (<10 mg/day or ≥10 mg/day), and geographic region (North America, Latin America, Europe, Asia, Japan, Rest of World) in the model. The analysis will be based on the mITT population and missing data will be handled using NRI. P-values from the Fisher's exact test will also be reported as a sensitivity analysis, when logistic regression sample size requirements are not met (<5 subjects in any category for any factor).

As supplementary analyses,

• to determine the impact of important protocol deviations, the primary analysis detailed above will also be conducted on the per-protocol population



#### 6.15. Secondary Endpoints/Estimand Analyses

The secondary endpoints per composite estimand strategy (the primary estimand as described in Section 6.5.2) without violation of concomitant medication rules: (i) initiating or increasing in dose of corticosteroids, antimalarial, or immunosuppressant, or (ii) using prednisone >10 mg per day (or equivalent) after Week 12 are

- BICLA at Week 24
- SRI-4 at Week 24, and
- LLDAS at Week 24.

Under the composite estimand strategy, participants will be considered nonresponders at all subsequent visits after the first violation of concomitant medication rules regardless of their discontinuation status.

The analytical details specified in Section 6.14 will be followed. The supplementary analyses in Section 6.14 may also be considered for the secondary efficacy endpoints if deemed appropriate.

Description and derivation of secondary endpoints are described in a separate document, and the handling of missing data due to, for example, a missed visit is detailed in Appendix 1.







#### 6.19. Safety Analyses

All safety data will be descriptively summarized by treatment groups and analyzed based on the safety population. The safety population is defined as those patients who received at least 1 dose of study drug and did not discontinue the study for the reason "lost to follow-up" at the first postbaseline visit. The safety analyses include AEs, safety in special groups and circumstances, including adverse events of special interest, laboratory analytes, QIDS-SR16, C-SSRS, ECGs, and vital signs. The duration of exposure will also be summarized. The categorical safety measures will be summarized using IRs and analyzed by Fisher's exact test. The mean change in the continuous safety measures including vital signs, QIDS-SR16, physical characteristics, and laboratory values will be summarized by visits and analyzed by ANCOVA, with treatment and baseline values in the model. More details are provided in subsequent sections.





Not all displays described in this section will necessarily be included in the CSRs. Any display described and not provided in the CSR would be available upon request. Not all displays will necessarily be created as a "static" display. Some may be incorporated into interactive display tools instead of or in addition to a static display. Any display created interactively will be included in the CSR if deemed relevant to the discussion.

#### 6.19.1. Extent of Exposure

Duration of exposure to study drug will be summarized for the safety population by treatment group. Exposure will be calculated as the date of last dose of study drug (or date of discontinuation) minus the date of first dose of study drug plus 1 day. Total PYs of exposure will be reported for each treatment group for overall duration of exposure. Descriptive statistics (n, mean, SD, minimum, first quartile, median, third quartile, and maximum) will be provided for patient-days of exposure and the frequency of patients falling into different exposure ranges will be summarized. Exposure ranges are as follows:

- $\geq$ 4 weeks,  $\geq$ 12 weeks, and  $\geq$ 24 weeks
- >0 to <4 weeks,  $\ge 4$  weeks to <12 weeks,  $\ge 12$  weeks to <24 weeks, and  $\ge 24$  weeks

Overall exposure will be summarized in total PYs, which are calculated according to the following:

Exposure in PYs = sum of duration of exposure in days (for all patients in treatment group) / 365.25

No p-values will be reported in these tables as they are intended to describe the characteristics of the study sets.

#### 6.19.2. Adverse Events

#### 6.19.2.1. Adverse Events

AEs are recorded in the eCRF. Each AE will be coded to SOC and PT, using the MedDRA version that is current at the time of database lock. Severity of AEs is recorded as mild, moderate, or severe.

TEAEs are defined as events that either first occurred or worsened in severity after the first dose of study drug and the earliest of the visit study drug disposition date or the last visit date during the treatment period, whichever occurred first, and up to 30 days after study treatment discontinuation. The MedDRA LLT will be used in defining which events are treatment-emergent. The maximum severity for each LLT during the baseline period until the first dose of the study medication will be used as baseline. If an event is preexisting during the baseline period, but it has missing severity, and the event persists during the treatment period or up to 30 days after treatment discontinuation, then the baseline severity will be considered mild for
determining any postbaseline treatment-emergence (that is, the event is treatment-emergent unless the severity is coded mild at postbaseline). If an event occurring postbaseline has a missing severity rating, then the event is considered treatment-emergent. Should there be insufficient data for an AE start date to make this comparison (for example, the AE start year is the same as the treatment start year, but the AE start month and day are missing), the AE will be considered treatment-emergent. For events occurring on the day of the first dose of study treatment, the day and time of the onset of the event will both be used to distinguish between pretreatment and posttreatment in order to derive treatment-emergence.

In general, summaries will include the number of patients in the safety population (N), frequency of patients experiencing the event (n), and relative frequency (that is, percentage; n/N\*100).

In an AE overview table, the number and percentage of patients in the safety analysis set who experienced death, an SAE, any TEAE, permanent discontinuation from study drug due to an AE, temporary interruption of study drug due to an AE or laboratory abnormality, or a severe TEAE will be summarized by treatment group.

The number and percentage of patients with TEAEs will be summarized by treatment group in 2 formats listed below. For events that are gender specific, the denominator and computation of the percentage will only include patients from the given gender.

- by MedDRA PT nested within SOC with SOCs ordered alphabetically, and events ordered within each SOC by decreasing frequency in the LY3471851
- by MedDRA PT with events ordered by decreasing frequency in the LY3471851 treatment group.

AEs leading to permanent discontinuation of study drug and AEs leading to temporary interruption of study drug will also be summarized by treatment group using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC in the LY3471851 treatment group.



The number and percentage of patients with TEAEs will be summarized by maximum severity by treatment using MedDRA PT ordered by decreasing frequency for the common TEAEs. For each patient and TEAE, the maximum severity for the MedDRA level being displayed is the

maximum postbaseline severity observed from all associated LLTs mapping to that MedDRA PT.

#### 6.19.2.2. Serious Adverse Events

An individual listing of all AEs including preexisting conditions will be provided. A separate listing will include AEs that led to permanent discontinuation from the study drug. In addition, a listing of AEs that occur more than 30 days after study treatment discontinuation will be provided.

With the ICH E2A guideline, a SAE is any AE that results in 1 of the following outcomes:

- death
- initial or prolonged inpatient hospitalization
- a life-threating experience (that is, immediate risk of dying)
- persistent or significant disability/incapacity
- congenital anomaly/birth defect, or
- considered significant by the investigator for any other reason.

The number and percentage of patients who experienced any ICH-defined SAE will be summarized by treatment group during the treatment and follow-up periods using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC in the LY3471851 cells treatment group. In addition, the SAEs will be summarized by treatment group using MedDRA PT without SOC. An individual listing of all SAEs will be provided.







#### 6.19.3.3. Malignancies

Malignancies will be identified using terms from the Malignant tumors SMQ (SMQ 20000194). Malignancies excluding NMSC and NMSC will be reported separately.

A listing including all malignancy cases will be provided. An NMSC flag will be provided using the following MedDRA PTs (the list will be updated depending on the MedDRA version used for analysis):

- Squamous cell carcinoma of skin (10041834)
- Bowen's disease (10006059)
- Basal cell carcinoma (10004146)
- Basosquamous carcinoma (10004178)
- Basosquamous carcinoma of skin (10004179)
- Squamous cell carcinoma (10041823)
- Skin squamous cell carcinoma metastatic (10077314)
- Skin cancer (10040808), and
- Carcinoma in situ of skin (10007390).

The number and percentage of patients with TEAE-associated malignancies excluding NMSC and NMSC will be summarized by treatment group. In addition, the IR (for detail, see Section 6.19) and 95% CI will be calculated for the overall observation time. All cases identified by Malignant tumors SMQ will be assessed after database lock by the medical team to determine (1) confirmed NMSC cases and (2) symptom and date that triggered the malignancy investigation or diagnosis. An additional listing based on medical review may also be provided if deemed necessary. All cases reported in the study database or by Lilly Safety System report, disregarding the length of gap between the last treatment dose date and the event date will be included.

# 6.19.4. Injection Site Reaction

At every visit following the first dose and prior to any blinded study activity, an independent ISR assessor who is not involved with other study procedures will evaluate each participant for the presence of ISRs between the visits.

The number and percentage of patients who experienced an ISR will be summarized by treatment group and by visit. The number and percentage of patients with the following ISR records will be summarized by treatment group and by visit. Details about ISR records are referred to the case report form.

- anatomical location of the injection site reaction
- abdomen side
- directionality of the anatomical location of the administration
- arm side
- thigh side
- whether the subject have any injection site erythema (reddening) or not
- severity of the injection site erythema
- whether the subject have any injection site induration (hardening or thickening of tissue) or not
- severity of the injection site induration
- whether the subject have any injection site pain (including burning) or not

- severity of the injection site pain
- whether the subject have any injection site pruritus
- severity of the injection site pruritus
- whether the subject have any injection site edema (swelling or accumulation of fluid in tissues at height above normal skin) or not
- severity of the injection site edema, and
- when did the injection related event occur, in relationship to the study treatment.

The frequency of the maximum severity of ISRs will be summarized by treatment group.



if the planned sample size is not achieved due to an insufficient number of consenting and eligible participants.

## 6.19.5. Clinical Laboratory Evaluation

All laboratory tests will be presented using the Système International of units (SI) and conventional (CN) units. For topics of safety in special groups and circumstances, laboratory test units will be specified for each analysis.

Lilly LCTPB reference limits will be used to define the low and high limits because it is generally desirable for limits used for analyses to have greater specificity (identify fewer false positive cases) than reference limits used for individual patient management. When Lilly LCTPB reference ranges are unavailable, then central laboratory (Covance) reference ranges will be used. For the 4 key hepatic laboratory assessments (ALT, AST, total bilirubin, and ALP), central laboratory reference ranges (Covance) will be used and all results pertaining to these assessments will be included as a separate analysis to address the risk of liver injury as a special safety topic (see Section 6.19.5.1). Central laboratory reference ranges (Covance) will also be used to evaluate immunoglobulins and lymphocyte cell subsets (see Sections 6.19.5.3 and 6.19.5.7). See Appendix 6 for details of the reference range by laboratory analytes.

The LDL/HDL ratio will be derived as the ratio of LDL cholesterol to HDL cholesterol. There are no Lilly LCTPB reference ranges or central lab reference ranges for the LDL/HDL ratio.

The following will be conducted for laboratory analyte measurements collected quantitatively:

- Box plots for observed values: Values at each visit (starting at randomization) and change from baseline to each visit and to last postbaseline measure will be displayed in box plots for patients who have a baseline and at least 1 postbaseline visit. For visits included in the treatment period, patients will be included only if the visit occurs on or before the date of treatment discontinuation/completion. Follow-up visit will be the first visit that occurred during the Follow-up period. Individual measurements outside of reference limits will also be displayed using distinct symbols overlaying the box plot. Original-scale data will be used for the display but for some analytes (for example, immunoglobulins) a logarithmic scale will be used to aid in viewing the measures of central tendency and dispersion. Unplanned measurements will be excluded. Descriptive summary statistics will be included in a table below the box plot. These box plots will be used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries. A p-value for change from baseline to endpoint will be provided using an ANCOVA model with explanatory term for treatment and the baseline value as a covariate. Endpoint will be the last observation where patient is on treatment.
- Treatment-emergent high/low analyses: the number and percentage of patients with treatment-emergent high and low laboratory results at any time will be summarized by treatment group. Planned and unplanned measurements will be included. A treatment-emergent high result is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time during the treatment period and up to 60 days after treatment discontinuation. A treatment-emergent low result is defined as a change from a value greater than or equal to the low limit at all baseline visits to a value less than the low limit at any time during the treatment period and up to 60 days after treatment discontinuation. The Fisher's exact test will be used for the treatment comparisons.

A listing of abnormal findings will be provided. The listing will include, but not be limited to, patient ID, treatment group, laboratory collection date, analyte name, and analyte finding.

#### 6.19.5.1. Abnormal Hepatic Tests

Analyses for abnormal hepatic tests involve 4 laboratory analytes: ALT, AST, total bilirubin, and ALP. Analyses for the change from baseline to last visit that occurred on or before the date of treatment discontinuation and shift tables are described in Section 6.19.5. This section describes additional analyses for the topic. The central laboratory reference ranges (Covance) will be used for ALT, AST, total bilirubin, and ALP hepatic laboratory assessments.

The number and percentage of patients with the following abnormal elevations in hepatic laboratory tests at any time up to 60 days after treatment discontinuation will be summarized by treatment group. LY3471851 groups will be compared to placebo using Fisher's exact text:

- The percentages of patients with an ALT measurement ≥3×, 5×, and 10× the central laboratory ULN during the treatment and follow-up periods will be summarized for all patients with a postbaseline value and for subsets based on various levels of baseline.
  - O The analysis of  $3 \times$  ULN will contain 4 subsets: patients whose nonmissing maximum baseline value is  $\leq 1 \times$  ULN; patients whose maximum baseline is  $\geq 1 \times$  ULN, but  $\leq 3 \times$  ULN; patients whose maximum baseline value is  $\geq 3 \times$  ULN; and patients whose baseline values are missing.
  - o The analysis of 5× ULN will contain 5 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN; patients whose maximum baseline is >1× ULN, but <3× ULN; patients whose maximum baseline is ≥3× ULN, but <5× ULN; patients whose maximum baseline value is ≥5× ULN; and patients whose baseline values are missing.</p>
  - o The analysis of 10× ULN will contain 6 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN; patients whose maximum baseline is >1× ULN, but <3× ULN; patients whose maximum baseline is ≥3× ULN, but <5× ULN; patients whose maximum baseline is ≥5× ULN, but <10× ULN; patients whose maximum baseline value is ≥10× ULN; and patients whose baseline values are missing.
- The percentages of patients with an AST measurement greater than or equal to 3×, 5×, and 10× the central laboratory ULN during the treatment and follow-up periods will be summarized for all patients with a postbaseline value and for subsets based on various levels of baseline. Analyses will be constructed as described above for ALT.
- The percentages of patients with a total bilirubin measurement greater than or equal to 2 × the central laboratory ULN during the treatment period will be summarized for all patients with a postbaseline value and subset into 4 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN; patients whose maximum baseline is >1× ULN but < 2× ULN; patients whose maximum baseline value is ≥2× ULN; and patients whose baseline values are missing.
- The percentages of patients with an ALP measurement ≥1.5× the central laboratory ULN during the treatment and follow-up periods will be summarized for all patients with a postbaseline value and subset into 4 subsets: patients whose nonmissing maximum baseline value is ≤1× ULN; patients whose maximum baseline is >1× ULN but <1.5× ULN; patients whose maximum baseline value is ≥1.5× ULN; and patients whose baseline values are missing.

Second, to further evaluate potential hepatotoxicity, an eDISH plot will be created for all patients whether treated with LY3471851 and/or other treatment using the whole study and follow-up periods. Each patient with at least 1 postbaseline ALT and total bilirubin will be included in the eDISH. The points correspond to maximum total bilirubin and maximum ALT, even if not

obtained from the same blood draw. A listing of patients potentially meeting Hy's rule will be provided (defined as greater than or equal to  $3 \times$  ULN for ALT or AST, and greater than or equal to  $2 \times$  ULN for total bilirubin, not necessarily at the same time).

Third, a listing will be provided to the medical safety team for internal review according to the following SMQs:

- broad and narrow terms in the Liver-related investigations, signs and symptoms SMQ (SMQ 20000008)
- broad and narrow terms in the Cholestasis and jaundice of hepatic origin SMQ (SMQ 20000009)
- broad and narrow terms in the Hepatitis non-infectious SMQ (SMQ 20000010)
- broad and narrow terms in the Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions SMQ (SMQ 20000013), and
- narrow terms in the Liver-related coagulation and bleeding disturbances SMQ (SMQ 20000015)

### 6.19.5.2. Hematologic Changes

Hematologic changes will be defined based on clinical laboratory assessments. CLASI will be applied for laboratory tests potentially related to myelosuppressive events (refer to Appendix 7).

Treatment-emergent laboratory abnormalities potentially related to myelosuppression occurring at any time during the treatment and follow-up periods and shift tables of baseline to maximum grade during the treatment and follow-up periods will be tabulated. Planned and unplanned measurements will be included. Treatment emergence will be characterized using the following 5 criteria (as appropriate to the grading scheme):

- any increase in postbaseline CTCAE grade from worst baseline grade
- increase to Grade 1 or above at worst postbaseline
- increase to Grade 2 or above at worst postbaseline
- increase to Grade 3 or above at worst postbaseline, and
- increase to Grade 4 at worst postbaseline.

Shift tables will show the number and percentage of patients based on baseline to maximum during the treatment and follow-up periods, with baseline depicted by the most extreme grade during the baseline period. With each shift table, a shift table summary displaying the number and percentage of patients with maximum postbaseline results will be presented by treatment group for each treatment period within the following categories:

- decreased; post-baseline category < baseline category
- increased; post-baseline category > baseline category, and
- same; postbaseline category = baseline category.

A laboratory-based treatment-emergent outcome related to increased platelet count will be summarized in a similar fashion. Treatment-emergent thrombocytosis as a laboratory-based abnormality will be defined as an increase in platelet count from a maximum baseline value  $\leq$ 600 billion/L to any postbaseline value  $\geq$ 600 billion/L. Planned and unplanned measurements

will be included. A listing of patients with treatment-emergent thrombocytosis will be provided for safety review.



#### 6.19.5.4. Lipids Effects

Analyses for the change from baseline to last observation, and shift tables in total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides are described in Section 6.19.5.

TEAEs potentially related to hyperlipidemia will also be analyzed, based on reported AEs. The target surveillance term "Hyperlipidemia" is a Lilly-defined MedDRA search criteria list that is a subset of the PTs in the MedDRA SMQ "Dyslipidemia" that are related to elevated or increased lipids. MedDRA PTs, each with a narrow scope from the SMQ, for the target surveillance term are shown in Appendix 5. Frequency and relative frequency for each PT will be provided, ordered by decreasing frequency in the LY3471851

#### 6.19.5.5. Renal Function Effects

Effects on renal function will be assessed through analyses of creatinine, which are described in Section 6.19.5.

#### 6.19.5.6. Elevations in Creatine Phosphokinase

Analyses of creatine phosphokinase are described in Section 6.19.5.



## 6.19.6. Vital Signs and Other Physical Findings

Vital signs and physical characteristics include systolic blood pressure, diastolic blood pressure, pulse, weight, body mass index, and body temperature. Original-scale data will be analyzed. When these parameters are analyzed as continuous numerical variables, unplanned measurements will be excluded. When these parameters are analyzed as categorical outcomes, planned and unplanned measurements will be included.

The planned analyses described for the laboratory analytes in Section 6.19.5 will be used to analyze the vital signs and physical characteristics.

Table KFAJ.6.1 defines the low and high baseline values as well as the criteria used to define treatment-emergence based on postbaseline values. Postbaseline values include all values after baseline in the treatment and follow-up periods. The blood pressure and pulse rate criteria are consistent with the document *Selected Reference Limits for Blood Pressure, Orthostasis, and ECG Numerical Parameters (Including Heart Rate) for Use in Phase II-IV Clinical Trials Version 1.1* approved on 8 March 2013 as recommended by the Lilly Cardiovascular Safety Advisory Committee.

Table KFAJ.6.1. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure and Pulse Measurement, and Categorical Criteria for Weight Changes for Adults

| Parameter | | |
|---|---|---|
| (Units of Measure) | Low | High |
| Systolic Blood Pressure | ≤90 (low limit) and decrease from | ≥140 (high limit) and increase from highest |
| (mm Hg) | lowest value during baseline ≥20 if | value during baseline ≥20 if <140 at each |
| | >90 at each baseline visit | baseline visit |
| Diastolic Blood Pressure | ≤50 (low limit) and decrease from | ≥90 (high limit) and increase from highest |
| (mm Hg) | lowest value during baseline ≥10 if | value during baseline ≥10 if <90 at each |
| | >50 at each baseline visit | baseline visit |
| Pulse | <50 (low limit) and decrease from | >100 (high limit) and increase from highest |
| (beats per minute) | lowest value during baseline ≥15 if | value during baseline ≥15 if ≤100 at each |
| | ≥50 at each baseline visit | baseline visit |
| Weight | (Loss) decrease ≥7% from lowest | (Gain) increase ≥7% from highest value |
| (kilograms) | value during baseline | during baseline |

Abbreviation: mm Hg = millimeters of mercury.

# 6.19.7. Additional Safety Sections

#### 6.19.7.1. Symptoms of Depression (QIDS-SR16)

The QIDS-SR16 is a 16-item, self-report instrument intended to assess the existence and severity of symptoms of depression as listed in the American Psychiatric Association's *Diagnostic and Statistical Manual of Mental Disorders*, 4th Edition (DSM-IV; APA 1994). Patients are asked to consider each statement as it relates to the way they have felt for the past 7 days. There is a unique 4-point ordinal scale for each item with scores ranging from 0 to 3 reflecting increasing depressive symptoms as the item score increases. Additional information and the QIDS-SR16 questions may be found on the University of Pittsburgh Epidemiology Data Center website (http://www.ids-qids.org/index.html). A key reference for this instrument covers its psychometric properties for use in patients with chronic major depression (Rush et al. 2003). Quick Inventory of Depressive Symptomatology was developed at UT Southwestern.

The QIDS-SR16 total score is derived as the sum of the scores across the 9 scale domains. For scale domains that contain more than 1 item, the domain score is the highest item rating given across the items within that domain:

- sleep: the highest score on any 1 of the 4 sleep items (items 1 to 4)
- depressed mood: Item 5
- weight/appetite change: the highest score on any 1 of the 4 weight items (items 6 to 9)
- psychomotor changes: the highest score on either of the 2 psychomotor items (items 15 and 16)
- concentration: item 10
- worthlessness/Guilt: item 11
- suicidal ideation: item 12
- decreased interest: item 13, and
- decreased energy: item 14.

In the presence of missing data, the following rules will be employed to derive the total score. Firstly, considering the 3 multi-item domains (sleep, weight/appetite change, psychomotor changes), the domain score should be based on the maximum value across the appropriate items, and it should be missing only if each item is missing. Further, considering the 9 domain scores, the total score should be derived as missing if there are 3 or more domains that are missing; if 1 or 2 domain scores are missing, then the total score should be derived using a total score that is prorated to the full scale range (0 to 27) based on the available domain scores, retaining 1 decimal place in the total score derived in the presence of missing data.

The QIDS-SR16 total scores will also be categorized in the following severity classes as shown in Table KFAJ.6.3.

Table KFAJ.6.3. QIDS-SR16 Severity of Depressive Symptoms Categories Based on the QIDS-SR16 Total Score

| QIDS-SR16 Severity of Depressive Symp | toms |
|---------------------------------------|-----------------------|
| Category | QIDS-SR16 Total Score |
| 0 = None | 0-5 |
| 1 = Mild | 6-10 |
| 2 = Moderate | 11-15 |
| 3 = Severe | 16-20 |
| 4 = Very Severe | 21-27 |

Abbreviation: QIDS-SR16 = Quick Inventory of Depressive Symptomatology Self-Rated.

Treatment differences in mean change QIDS-SR16 total score will be analyzed using the MMRM model described in Section 6.2. Only visits that occur on or before the date the patient discontinued treatment will be included in this analysis.

Using the QIDS-SR16 Severity of Depressive Symptoms Categories shown in Table KFAJ.6.3, shift tables will show the number and percentage of patients with total score in each category based on baseline to maximum category during the treatment period and up to 60 days after treatment discontinuation, with baseline depicted by the most extreme category during the baseline period, with further summarization of change from baseline in severity using categories of any improvement, no change, and any worsening, by treatment. Similarly, shift tables will be created for the QIDS-SR16 suicidal ideation item (Item 12) responses.

Treatment-emergent changes in QIDS-SR16 total score severity categories will be characterized as follows:

- Increase (from None) to Mild, Moderate, Severe, or Very Severe
- Increase (from None or Mild) to Moderate, Severe, or Very Severe
- Increase (from None, Mild, or Moderate) to Severe or Very Severe
- Increase (from None, Mild, Moderate, or Severe) to Very Severe

Treatment-emergent changes in QIDS-SR16 suicidal ideation item (Item 12) responses will be characterized as follows:

- Increase (from 0) to 1 to 3
- Increase (from 0 to 1) to 2 to 3, and
- Increase (from 0 to 2) to 3.

#### 6.19.7.2. Columbia Suicide Severity Rating Scale

Suicidal ideation, suicidal behavior, and self-injurious behavior without suicidal intent, based on the C-SSRS, will be listed by patient and visit. Only patients that show suicidal ideation/behavior or self-injurious behavior without suicidal intent will be displayed (that is, if a patient's answers are all 'no' for the C-SSRS, then that patient will not be displayed). However, if a patient reported any suicidal ideation/ behavior or self-injurious behavior without suicidal intent at any time point then all their ideation and behavior will be displayed, even if not positive.

## 6.20. Other Analyses

## 6.20.1. Subgroup Analyses

Subgroup analysis will be conducted on SLEDAI-4 and SRI-4 at Week 24 with the composite estimand strategy based on the mITT population. Subgroup analysis may be conducted on BICLA at Week 24 with the composite estimand strategy for mITT population with at least 1 baseline BILAG A score or 2 baseline BILAG B scores. Missing data will be handled using NRI. Subgroups to be analyzed are listed in Section 6.7.1. Subgroup analyses on other efficacy endpoints may be performed as deemed appropriate.

Descriptive statistics will be provided for each treatment and stratum of a subgroup as outlined, regardless of sample size. Each categorical variable will be analyzed individually with a logistic model that contains the treatment, the subgroup variable, and subgroup by treatment interaction. The treatment-by-subgroup interaction will be tested at the 10% significance level to determine whether treatment differences are the same for each subgroup category. For the categorical variables, the number of responders and response rate will be reported for each subgroup.



# 6.20.3. Annual Report Analyses

Annual report analyses will be stated in a separate document.

# 6.20.4. Clinical Trial Registry Analyses

Additional analyses will be performed for the purpose of fulfilling the CTR requirements.

Analyses provided for the CTR requirements include the following:

Summary of AEs, provided as a dataset that will be converted to an XML file. Both SAEs and "other" AEs are summarized by treatment group, by MedDRA PT.

- An AE is considered "serious," whether or not it is a TEAE.
- An AE is considered in the "other" category if it is both a TEAE and is not serious. For each SAE and "other" AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term, and
  - o the number of events experienced



• AE reporting is consistent with other document disclosures for example, the CSR, manuscripts, and so forth.





# 6.22. Data Monitoring Committee

Not applicable. An IAC will be used to conduct the interim analysis.

Details of the planned interim data analyses and the assessment committee data review process are included in an assessment committee charter.

# 7. Unblinding Plan

A separate unblinding plan will be prepared.

#### 8. References

- American Psychiatric Association. *Diagnostic and Statistical Manual of Mental Disorders*. 4th ed. Arlington (VA): American Psychiatric Association; 1994.
- Andersen, Scott W, Millen BA. On the practical application of mixed effects models for repeated measures to clinical trial data. *Pharmaceutical statistics* 12.1 (2013): 7-16.
- Bretz F, Pinheiro JC, Branson M. Combining multiple comparisons and modeling techniques in dose-response studies. *Biometrics*. 2005;61(3):738-748. https://doi.org/ 10.1111/j.1541-0420.2005.00344.x
- [FDA] Food and Drug Administration. Office of Clinical Pharmacology Division of Pharmacometrics. Request for Qualification of MCP-Mod as an efficient statistical methodology for model-based design and analysis of Phase II dose finding studies under model uncertainty. 22 April 2015. Accessed December 09, 2022. https://www.fda.gov/media/99313/download
- Gould AL. BMA-Mod: A Bayesian model averaging strategy for determining dose-response relationships in the presence of model uncertainty. *Biom J.* 2019;61(5):1141-1159. https://doi.org/ 10.1002/bimj.201700211
- Rush AJ, Trivedi MH, Ibrahim HM, et al. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. *Biol Psychiatry*. 2003;54(5):573-583.

Winthrop KL, Novosad SA, Calabrese L, et al. Opportunistic infections and biologic therapies in immune-mediated inflammatory disease: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance. *Ann Rheum Dis*. 2015;74(12):2107-2116. https://doi.org/10.1136/annrheumdis-2015-207841.

# 9. Appendices

# Appendix 1. Description and Derivation of Efficacy Outcomes Measures and Endpoints

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| SLEDAI-2K | The SLEDAI-2K is a global disease activity instrument that focuses on high-impact disease manifestations across 9 organ domains: constitutional, mucocutaneous, musculoskeletal, vascular, cardiorespiratory, central nervous system, immunologic, renal, and hematologic. | SLEDAI-2K<br>Total Score | Calculated by summing the weighted organ manifestation. | Any item scores are missing (not done, not assessed, NA or empty), but the visit occurred. • Baseline data for that item can be carried forward from the last non-missing data during the screening period. • Postbaseline data for that item can be carried forward from the last non-missing data if that data is obtained within the previous 34 days of that visit. After imputation, • If any item is still missing at the baseline visit, it will be imputed as 0. • For Renal domain, if urinary casts, hematuria and pyuria items are still missing for any post-baseline visit, they will be imputed as 0. |
| | | Individual Organ Domain Improvement Defined by SLEDAI-2K | Patients with SLEDAI-2K score >0 within the organ domain at baseline, and able to decrease SLEDAI-2K (from baseline) within each organ domain score, separately. | Missing if any SLEDAI-2K item for that organ domain remains missing after instrument level imputation rules are applied. |
| | | Individual Organ Domain No Worsening Defined by SLEDAI-2K | Among patients with at least one SLEDAI-2K item = 0 (not present) in the organ domain score at baseline, no increment of SLEDAI-2K organ domain score from baseline within each organ domain score, separately. | Missing if any SLEDAI-2K item for that organ domain remains missing after instrument level imputation rules are applied. |

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| | | No worsening<br>from baseline<br>in SLEDAI-2K | No increment from baseline of >0 points in SLEDAI-2K | Missing if any SLEDAI-2K item for<br>that organ domain remains missing<br>after instrument level imputation rules<br>are applied. |
| SLEDAI-4 | SLEDAI-4 is an index to<br>measure overall<br>improvement in disease<br>activity (SLEDAI-2K) | SLEDAI-4<br>Responder | A ≥4-point reduction in SLEDAI-2K score from baseline. | Missing if SLEDAI-2K total score is missing after instrument level imputation rules are applied. |
| SRI-4 | SRI-4 is a composite index to<br>measure overall<br>improvement in disease<br>activity (SLEDAI-2K) while<br>ensuring there is no<br>worsening in other organ<br>systems (BILAG and PGA) | SLE Responder<br>Index 4 | <ul> <li>A decrease in SLEDAI-2K ≥4 (from baseline)</li> <li>No new BILAG A and no more than 1 new BILAG B disease activity score / organ domain (both compared with baseline), and</li> <li>No worsening in PGA (defined as an increase of 0.3 points [10 mm] from baseline)</li> </ul> | After each instrument level imputation rule is applied and there is still at least one missing component, • if the nonmissing components are all 'Y' then SRI-4 is missing. • if any of the nonmissing component is 'N' then the SRI-4 is 'N.' |
| BILAG-2004 | BILAG2004 assesses 97 clinical signs, symptoms and laboratory parameters across 9 organ system domains: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal and hematological | BILAG | A, B, C, D, or E score will be used in analyses for each of the 9 individual organ systems. | Within each organ domain (except renal and hematological), any missing data will be assumed to be 'Not present' if there is at least 1 nonmissing item in that organ. If all items in one organ domain are completely missing but the visit occurred, then the letter score of that organ from the previous visit will be pulled forward, provided data were obtained within 34 days of visit; otherwise missing except when the letter score from the last nonmissing visit is E, then E score will be pulled forward. For the renal and hematological domains, |

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| | | | | <ul> <li>If all item within this domain is 'NA', then items are coded as 'No.'</li> <li>If any vital/lab item with "Yes" but vital and lab value is missing, then vital/lab values will be pulled forward from scheduled and unscheduled post-baseline visits, provided data were obtained within 34 days of visit; otherwise missing.</li> <li>If all items in one organ domain are completely missing not 'NA' but the visit occurred, then the letter score of that organ from the previous visit will be pulled forward, provided data were obtained within 34 days of visit; otherwise missing except when the letter score from the last non-missing visit is E, then E score will be pulled forward.</li> </ul> |
| | | BILAG improvement | <ul> <li>Reduction of all baseline BILAG A to B/C/D and baseline BILAG B to C/D</li> <li>No BILAG worsening in other organ systems, where worsening is defined as ≥1 new BILAG A or ≥2 new BILAG B</li> </ul> | For the reduction part, missing if any of 9 domains at baseline or at the visit remains missing after instrument level imputation rules are applied except when the missing is at the baseline (any one or all domains) and the value at the visit is not A or B, then the other non-missing organ domains will be used to determine the response status. |

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| | | No BILAG<br>worsening | No new BILAG A and no more than 1 new BILAG B disease activity score (both compared with baseline), where worsening is defined as ≥1 new BILAG A or ≥2 new BILAG B, both compared with the baseline. The baseline BILAG A improved to BILAG B at the visit will not be considered as the new BILAG B. | For the no worsening part, Missing if any of 9 domains at baseline or at the visit remains missing after instrument level imputation rules are applied except when the baseline (any one or all domains) is BILAG A and the value at the visit is missing, then the other non-missing organ domains will be used to determine the response status. If both components are missing or one component is missing and the other one is 'Y,' then missing. If at least one component is 'N', then 'N.' Missing if any of 9 domains at baseline or at the visit remains missing after instrument level imputation rules are applied except when the baseline (any one or all domains) is BILAG A and the value at the visit is missing, then the other nonmissing organ domains will be used to determine the response status. |
| | | Individual<br>Organ Domain | Among patients with BILAG A or B at baseline and able to reduce the baseline BILAG A to | Missing if baseline or value remains missing after instrument level |
| | | Improvement | B/C/D and BILAG B to C/D for each organ | imputation rules are applied. |
| | | Defined by | domain, separately. | 1 |
| rd. | 8 | BILAG | 70.1 | |

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| | | Individual Organ Domain No Worsening Defined by BILAG | Among patients without BILAG A at baseline, no increment of baseline BILAG B/C/D/E to A and baseline BILAG C/D/E to B for each organ domain, separately. | Missing if baseline or value remains missing after instrument level imputation rules are applied. |
| PGA | The PGA is the physician's assessment of the patient's overall disease activity due to SLE. It is scored using a visual analog scale where | PGA score<br>PGA category | Permitted range of values is from 0 to 100 mm. PGA categories are defined as: None (0) = '0 mm', Mild (>0 and <1.5) = '>0 to < 50 mm', Moderate ( $\ge$ 1.5 to $\le$ 2.5) = ' $\ge$ 50 mm to $\le$ 83mm', Severe (>2.5) = '>83mm'. | If the visit occurred, data can be carried forward if obtained within 34 days of visit; otherwise missing. |
| | 0 mm indicates no disease<br>activity and 100 mm<br>indicates the most severe<br>disease activity possible.<br>There are benchmarks of 0 | No worsening in PGA | Worsening is defined as an increase of ≥0.3 points (10 mm) from baseline. Therefore, no worsening is defined as any decrease, no change, or <0.3 points (10 mm) increase from baseline. | Missing if baseline or value remains missing after instrument level imputation rules are applied. |
| | (0 mm), 1 (33 mm), 2<br>(67 mm), and 3 (100 mm) on<br>the line corresponding to no,<br>mild, moderate, and severe<br>SLE disease activity,<br>respectively. | PGA ≤1 | PGA ≤33 mm | Missing if value remains missing at the visit after instrument level imputation rules are applied. |
| BICLA | BICLA is a composite index<br>to measure overall<br>improvement in disease<br>activity (BILAG) while<br>ensuring there is no<br>worsening in other organ<br>systems (SLEDAI and PGA) | BILAG Based<br>Composite<br>Lupus<br>Assessment | BILAG Improvement Reduction of all baseline BILAG A to B/C/D and baseline BILAG B to C/D No BILAG worsening in other organ systems, where worsening is defined as ≥1 new BILAG A or ≥2 New BILAG B No worsening from baseline in SLEDAI- 2K, where worsening is defined as an increase of >0 points from baseline in SLEDAI-2K | After each instrument level imputation rule is applied and there is at least one component missing, if the non-missing components are all 'Y' then BICLA will be missing. If any of the non-missing component is 'N' then the BICLA is 'N.' |

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| | | | No worsening from baseline in participants' lupus disease activity, where worsening is defined by an increase ≥0.30 points on a 3-point PGA VAS. | |
| LLDAS | The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. | LLDAS | <ul> <li>SLEDAI-2K ≤ 4, with no activity in SLEDAI-2K major organ systems (CNS, Vascular, Renal, Cardiorespiratory and Constitutional), where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0.</li> <li>No new features of Lupus disease activity in SLEDAI-2K compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0.</li> <li>PGA ≤1</li> <li>Current prednisone or equivalent ≤7.5 mg/day</li> </ul> | After each instrument level imputation rule is applied and there is at least one component missing, if the non-missing components are all 'Y' then LLDAS will be missing. If any of the nonmissing component is 'N' then the LLDAS is 'N.' |

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| SLEDAI | The SFI uses the SLEDAI | SFI Flare | No derivation; used as entered. | The absence of a flare record, or 'Non |
| Flare Index | score, disease activity | | | Applicable,' both are indicative of no |
| | scenarios, treatment changes, | , | | occurrence of flare. |
| | and PGA to define | Time to first | Time to first flare will be derived as the first | Not applicable |
| | mild/moderate and severe | flare | date of most recent flare minus date of first | |
| | flares. | | injection plus 1. | |









Abbreviations: ACR = American College of Rheumatology; BICLA = British Isles Lupus Assessment Group-based Composite Lupus Assessment; BILAG =
British Isles Lupus Assessment Group - 2004; CCI

CNS = central nervous system;

LLDAS = Lupus Low Disease Activity State; N = no; PGA = Physician
Global Assessment; Q2W = every 2 weeks; SFI = Self-Report Family Instrument; SLE = systemic lupus erythematosus; SLEDAI-2K = Systemic Lupus
Erythematosus Disease Activity Index 2000; SLEDAI-4 = a ≥4-point reduction in SLEDAI-2K score from baseline;

SRI-4 = Systemic Lupus Erythematosus Responder Index-4; VAS = Visual Analog Scale; Y = yes.

# **Appendix 2. Description of Efficacy Analyses**

The table below provides the detailed analyses including estimand strategy, analysis method, missing data imputation, analysis population, and analysis type.

| Measure | Endpoint | Estimand<br>Strategy | Analysis<br>Population | Comparison/<br>Timepoint | Analysis Method | Analysis Type |
|---|---|---|---|---|---|---|
| SLEDAI | SLEDAI-4 | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 – Primary<br>Other – Exploratory |
| | | Composite | Per-Protocol | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with NRI;<br>Fisher's Exact Test with NRI | Exploratory |
| | | Treatment<br>Policy | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | No worsening from<br>baseline in<br>SLEDAI-2K | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | SLEDAI Change from Baseline | Hypothetical | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | MMRM | Exploratory |
| | | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | MMRM with BOCF | Exploratory |
| | Individual Organ Domain Improvement Defined by SLEDAI-2K | Composite | mITT – Patients<br>with SLEDAI-2K<br>score > 0 within the<br>organ domain at<br>baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | Individual Organ<br>Domain Worsening<br>Defined by<br>SLEDAI-2K | Composite | mITT – Patients with at least one baseline SLEDAI- 2K = 0 in the organ domain at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |

| Measure | Endpoint | Estimand<br>Strategy | Analysis<br>Population | Comparison/<br>Timepoint | Analysis Method | Analysis Type |
|---|---|---|---|---|---|---|
| | Resolution of<br>Arthritis and/or<br>Rash by SLEDAI-<br>2K Components | Composite | mITT – Patients<br>with SLEDAI-2K<br>arthritis and/or rash<br>'Present' at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory |
| SRI-4 | SRI-4 | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory |
| | | Composite | Per-Protocol | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with NRI;<br>Fisher's Exact Test with NRI | Exploratory |
| BICLA | BICLA | Composite | mITT – Patients with at least 1 BILAG A or 2 BILAG B scores at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory |
| | | Composite | Per-Protocol – Patients with at least 1 BILAG A or 2 BILAG B scores at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Exploratory |
| LLDAS | LLDAS | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory |

| Measure | Endpoint | Estimand<br>Strategy | Analysis<br>Population | Comparison/<br>Timepoint | Analysis Method | Analysis Type |
|---|---|---|---|---|---|---|
| BILAG | BILAG<br>Improvement | Composite | mITT – Patients with at least 1 BILAG A or 2 BILAG B at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | BILAG No<br>Worsening | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | Individual Organ<br>Domain -<br>Improvement<br>Defined by BILAG | Composite | mITT – Patients<br>with BILAG A or B<br>within the organ<br>domain at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with NRI Fisher's Exact Test with NRI | Exploratory |
| | Individual Organ Domain - No Worsening Defined by BILAG | Composite | mITT – Patients with no BILAG A within the organ domain at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| PGA | PGA Change from<br>Baseline | Hypothetical | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | MMRM | Exploratory |

| Measure | Endpoint | Estimand<br>Strategy | Analysis<br>Population | Comparison/<br>Timepoint | Analysis Method | Analysis Type |
|---|---|---|---|---|---|---|
| | | Composite | mITT | LY3471851 vs Placebo at postbaseline visits in the treatment period | MMRM with BOCF | Exploratory |
| | No worsening in PGA | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | PGA ≤1 | Composite | mITT – Patients<br>with PGA > 1 at<br>baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |


















Abbreviations: Anti-dsDNA = anti-double stranded deoxyribonucleic acid; BICLA = British Isles Lupus Assessment Group-based Composite Lupus Assessment; BILAG = British Isles Lupus Assessment Group - 2004; BOCF = baseline observation carried forward; CCI

EACIT-Fatigue = Functional Assessment of Chronic Illness Therapy - Fatigue Scale: LLDAS =

FACIT-Fatigue = Functional Assessment of Chronic Illness Therapy – Fatigue Scale; LLDAS = Lupus Low Disease Activity State; mITT = modified intent-to-treat; MMRM = mixed models for repeated measures; NRI = nonresponder imputation; PGA = Physician Global Assessment; CCI

SF = Short Form;

SF-36 = 36-Item Short Form Health Survey; CCI

SLE = systemic lupus erythematosus; SLEDAI-2K = Systemic Lupus Erythematosus

Disease Activity Index 2000; SLEDAI-4 = a  $\geq$ 4-point reduction in SLEDAI-2K score from baseline; SLICC = Systemic Lupus Erythematosus International Collaborating Clinics; SRI-4 = Systemic Lupus Erythematosus Responder Index-4.

#### Appendix 3. Corticosteroid

All corticosteroid doses need to be converted to prednisone equivalent doses (as detailed in Section 6.9). If additional conversion factors are required, these will be added to the table below in a statistical analysis plan amendment prior to database lock.

The following table should be used for converting nonprednisone medications to prednisone equivalent:

Multiply the dose of the corticosteroid taken by the patient (in milligrams) in Column 1 by the conversion factor in Column 2 to get the equivalent dose of prednisone (in milligrams).

Example: Patient is taking 16 mg of methylprednisolone po daily. To convert to prednisone: 16 mg methylprednisolone  $\times$  1.25 = 20 mg prednisone. 16 mg of methylprednisolone po daily is equivalent to 20 mg of prednisone po daily.



## Appendix 4. List of MedDRA Preferred Terms for Potential Opportunistic Infections (POI)

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| Mycobacterial/ | Nocardiosis (II) | Nocardia sepsis | 10064952 | Narrow |
| Actino | | Nocardiosis | 10029444 | |
| | | Nocardia test positive | 10070131 | Broad |
| Mycobacterial/<br>Actino | - | Atypical mycobacterial infection | 10061663 | Narrow |
| | (II) | Atypical mycobacterial lower respiratory tract infection | 10075026 | |
| | | Atypical mycobacterial lymphadenitis | 10003755 | |
| | | Atypical mycobacterium pericarditis | 10055036 | |
| | | Atypical mycobacterial pneumonia | 10071075 | |
| | | Borderline leprosy | 10006029 | |
| | | Bovine tuberculosis | 10006049 | |
| | | Indeterminate leprosy | 10021700 | |
| | | Leprosy | 10024229 | |
| | | Lepromatous leprosy | 10024227 | |
| | | Mycobacterial infection | 10062207 | |
| | | Mycobacterial peritonitis | 10073514 | |
| | | Mycobacterium abscessus infection | 10064789 | |
| | | Mycobacterium avium complex immune restoration disease | 10058449 | |
| | | Mycobacterium avium complex infection | 10058806 | |
| | | Mycobacterium chelonae infection | 10071401 | |
| | | Mycobacterium fortuitum infection | 10049659 | |
| | | Mycobacterium kansasii infection | 10028447 | |
| | | Mycobacterium marinum infection | 10028452 | |
| | | Mycobacterium ulcerans infection | 10066289 | |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Superinfection<br>mycobacterial | 10075381 | |
| | | Tuberculoid leprosy | 10044729 | |
| | | Type 1 lepra reaction | 10070516 | |
| | | Type 2 lepra reaction | 10070517 | |
| | | Atypical mycobacterium test positive | 10070326 | Broad |
| | | Mycobacterial disease carrier | 10075025 | |
| | | Mycobacterium leprae test positive | 10070324 | |
| | | Mycobacterium test | 10070407 | |
| | | Mycobacterium test positive | 10070323 | |
| | | Ureaplasmal ulvovaginitis | 10081280 | |
| Mycobacterial/<br>Actino | Tuberculosis (I) | Adrenal gland tuberculosis | 10001358 | Narrow |
| | | Bone tuberculosis | 10056377 | |
| | | Choroid tubercles | 10008779 | |
| | | Congenital tuberculosis | 10010657 | |
| | | Conjunctivitis | 10010754 | |
| | | tuberculous | | |
| | | Cutaneous tuberculosis | 10011684 | |
| | | Disseminated Bacillus<br>Calmette-Guerin<br>infection | 10076666 | |
| | | Disseminated | 10013453 | |
| | | tuberculosis | | |
| | | Ear tuberculosis | 10014027 | |
| | | Epididymitis tuberculous | 10015004 | |
| | | Extrapulmonary tuberculosis | 10064445 | |
| | | Female genital tract tuberculosis | 10061150 | |
| | | Immune reconstitution inflammatory syndrome associated tuberculosis | 10072797 | |
| | | Intestinal tuberculosis | 10075268 | 7 |
| | | Joint tuberculosis | 10056367 | 7 |
| | | Lupus vulgaris | 10025143 | 7 |
| | | Lymph node tuberculosis | 10025183 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Male genital tract | 10061234 | |
| | | tuberculosis | | |
| | | Meningitis tuberculous | 10027259 | |
| | | Oesophageal | 10030200 | |
| | | tuberculosis | | |
| | | Oral tuberculosis | 10076879 | |
| | | Pericarditis tuberculous | 10055069 | 7 |
| | | Peritoneal tuberculosis | 10053583 | |
| | | Prostatitis tuberculous | 10064743 | |
| | | Pulmonary tuberculoma | 10066927 | |
| | | Pulmonary tuberculosis | 10037440 | |
| | | Renal tuberculosis | 10038534 | |
| | | Salpingitis tuberculous | 10039463 | |
| | | Silicotuberculosis | 10068876 | |
| | | Spleen tuberculosis | 10041640 | 7 |
| | | Thyroid tuberculosis | 10043774 | 7 |
| | | Tuberculoma of central | 10052883 | |
| | | nervous system | | |
| | | Tuberculosis | 10044755 | |
| | | Tuberculosis bladder | 10044758 | |
| | | Tuberculosis | 10061390 | |
| | | gastrointestinal | | _ |
| | | Tuberculosis liver | 10058120 | _ |
| | | Tuberculosis of central | 10061391 | |
| | | nervous system | 10044010 | _ |
| | | Tuberculosis of eye Tuberculosis of | 10044819<br>10044828 | $\dashv$ |
| | | genitourinary system | 10044828 | |
| | | Tuberculosis of | 10044846 | |
| | | intrathoracic lymph | 10011010 | |
| | | nodes | | |
| | | Tuberculosis of | 10044965 | |
| | | peripheral lymph nodes | | |
| | | Tuberculosis ureter | 10045026 | |
| | | Tuberculous abscess | 10052884 | |
| | | central nervous system | | |
| | | Tuberculous | 10071559 | |
| | | endometritis | | _ |
| | | Tuberculous laryngitis | 10045072 | |
| | | Tuberculous pleurisy | 10045104 | _ |
| | | Tuberculous | 10059161 | |
| | | tenosynovitis | 10072542 | Drand |
| | | Interferon gamma release assay | 10073542 | Broad |

| Interferon gamma release assay positive Mycobacterium tuberculosis complex test Mycobacterium tuberculosis complex test positive Tuberculin test false positive Tuberculin test false positive Tuberculin test false pagative Tuberculin test positive Tuberculin test Tuberculin | Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|---|
| Mycobacterium tuberculosis complex test | | | Interferon gamma | 10072866 | |
| Bacteria Bartonellosis Bacteria Bartonellosis Bacteria Bartonellosis 10003971 Narrow | | | release assay positive | | |
| test | | | Mycobacterium | 10070472 | |
| Mycobacterium tuberculosis complex test positive Tuberculid 10044725 Tuberculin test 10044726 Tuberculin test 10044726 Tuberculin test 10044726 Tuberculin test 10044726 Tuberculin test false negative Tuberculin test false 10074840 10044728 | | | tuberculosis complex | | |
| Bacteria Bartonellosis Tuberculin test 10044725 Tuberculin test 10044726 Tuberculin test 10044726 Tuberculin test 10074840 negative Tuberculin test false 10074840 negative Tuberculin test positive 10044728 Tuberculin test positive 10044728 Tuberculin test positive 10003971 Narrow Narrow Trench fever 10044582 Trench fever 10044582 Trench fever 10070157 Bartonella test positive 10070157 Bartonellosis 10004145 Cat scratch disease 10007729 Peliosis hepatis 10034229 Splenic peliosis 10068851 Tempylobacter sepsis 10070681 Narrow Campylobacter sepsis 10070681 Narrow Campylobacter 10007048 gastroenteritis Campylobacter 10007048 gastroenteritis Campylobacter test 10070025 Positive 10070025 Positive 10070025 Pontiac fever 10054161 Legionella test positive 10070092 Elisteria monocytogenes (invasive disease only) (II) Listeria sepsis 10063085 Listeria test 10075707 Broad Listeria test 10075707 Listeria test 10070094 Listeria test positive 10070094 Listeria sepositive 10070094 Listeria sepositive 10070094 Listeria test positive 10003271 Meningitis salmonella 100027254 Meningitis salmonella 10003271 Meningi | | | test | | |
| Lest positive | | | Mycobacterium | 10070325 | |
| Tuberculid | | | tuberculosis complex | | |
| Bacteria Bartonellosis (disseminated disease only) (V) Bartonellosis (disseminated disease only) (V) Bartonellosis (disseminated disease only) (V) Bartonella test 10075209 Broad Bartonella test 1007157 Bartonella test 10007157 Bartonella test 10007157 Bartonellosis 10004145 Cat scratch disease 10007729 Peliosis hepatis 10034229 Splenic peliosis 10068851 Campylobacter sepsis 1007688 Narrow Campylobacter colitis 10076769 Broad Campylobacter colitis 1007048 Broad Campylobacter test 1007048 Campylobacter test 1007048 Campylobacter test 10070025 Campylobacter test 10070025 Campylobacter test 10070025 Campylobacter test 10070025 Campylobacter test 10070016 Campylobacter test 10070016 Campylobacter test 10070025 Campylobacter test 10070016 Campylobacter test 10070025 Campylobacter test 10070025 Campylobacter test 10070016 Campylobacter 10070016 Campylobacter test 10070016 Campylobacter 10070016 Camp | | | - | | |
| Bacteria Bartonellosis (disseminated disease only) (V) Bartonellosis Bartonellosis (disseminated disease only) (V) Bartonella test 10075209 Broad Bartonellosis 10004145 Bartonella test 10075209 Broad Bartonellosis 10004145 Bartonellosis 10004145 Bartonellosis 10004145 Bartonellosis 10004145 Bartonellosis 10004145 Cat scratch disease 10007729 Peliosis hepatis 10034229 Splenic peliosis 10068851 Campylobacter iosis 10076769 Broad Campylobacter colitis 10076769 Broad Broad Campylobacter infection 10070048 Broad Campylobacter infection 10051226 Campylobacter test 10070025 positive Campylobacter infection 10061266 Narrow Pneumonia legionella 10035718 Pontiac fever 10054161 Legionella test 10070410 Broad Legionella test 10070092 Listeria encephalitis 10054116 Listeria test 10075707 Broad Listeria test 10070094 Listeria test 10070094 Listerioisis 10024641 Aortitis salmonella 10003271 Meningitis salmonella 10003271 Meningitis salmonella 100027254 Meningitis s | | | Tuberculid | 10044725 | |
| Bacteria Bartonellosis (disseminated disease only) (V) Bacillary angiomatosis 10003971 Narrow | | | Tuberculin test | 10044726 | |
| Bacteria Bartonellosis (disseminated disease only) (V) Bartonella test positive 10044728 Bacillary angiomatosis 10003971 Narrow | | | Tuberculin test false | 10074840 | |
| Bacteria Bartonellosis (disseminated disease only) (V) Trench fever 10044582 Bartonella test 10075209 Bartonella test 10070157 Bartonella test 10070157 Bartonella test 10070157 Bartonella test 10007157 Bartonella test 10007729 Peliosis hepatis 10034229 Splenic peliosis 10068851 Campylobacter sepsis 10070681 Narrow | | | | | |
| (disseminated disease only) (V) | | | Tuberculin test positive | 10044728 | |
| Only) (V) Bartonella test 10075209 Broad | Bacteria | | | 10003971 | Narrow |
| Bartonella test positive 10070157 | | | Trench fever | 10044582 | |
| Bartonellosis | | only) (V) | Bartonella test | 10075209 | Broad |
| Cat scratch disease 10007729 Peliosis hepatis 10034229 Splenic peliosis 10068851 Narrow | | | Bartonella test positive | 10070157 | |
| Peliosis hepatis 10034229 Splenic peliosis 10068851 | | | Bartonellosis | 10004145 | |
| Campylobacteriosis | | | Cat scratch disease | 10007729 | |
| Campylobacteriosis (invasive disease only) (V) Campylobacter sepsis 10070681 Narrow | | | Peliosis hepatis | 10034229 | |
| Campylobacter colitis 10076769 Broad | | | Splenic peliosis | 10068851 | |
| Campylobacter 10007048 gastroenteritis Campylobacter infection 10051226 Campylobacter test 10070025 positive Legionellosis (II) Legionella infection 10061266 Narrow Pneumonia legionella 10035718 Pontiac fever 10054161 Legionella test 10070410 Broad Legionella test 10070092 Listeria encephalitis 10054116 Narrow Listeria sepsis 10063085 (II) Meningitis listeria 10027248 Listeria test 10075707 Broad Listeria test 10070094 Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Arthritis salmonella 10074937 Narrow Arthritis salmonella 10003271 Meningitis salmonella 10007254 Narrow Arthritis salmonella 10007254 | | Campylobacteriosis | Campylobacter sepsis | 10070681 | Narrow |
| Campylobacter infection 10051226 Campylobacter test 10070025 positive | | (invasive disease only) | Campylobacter colitis | 10076769 | Broad |
| Campylobacter infection 10051226 Campylobacter test 10070025 positive | | (V) | Campylobacter | 10007048 | |
| Legionellosis (II) | | | gastroenteritis | | |
| Legionellosis (II) | | | Campylobacter infection | 10051226 | |
| Legionellosis (II) | | | | 10070025 | |
| Pneumonia legionella 10035718 Pontiac fever 10054161 Legionella test 10070410 Broad Legionella test positive 10070092 Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis 10054116 Narrow Listeria sepsis 10063085 Meningitis listeria 10027248 Listeria test 10075707 Broad Listeria test positive 10070094 Listeria test positive 10070094 Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Arthritis salmonella 10003271 Meningitis salmonella 100072254 Meningitis salmonella 10027254 | | T : 11 : (II) | • | 10061266 | NI |
| Pontiac fever | | Legionellosis (II) | | | Narrow |
| Legionella test 10070410 Broad | | | | | _ |
| Legionella test positive 10070092 | | | | | |
| Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis 10054116 Narrow | | | | | Broad |
| (invasive disease only) Listeria sepsis 10063085 (II) Meningitis listeria 10027248 Listeria test 10075707 Broad Listeria test positive 10070094 Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Aortitis salmonella 10074937 Arthritis salmonella 10003271 Meningitis salmonella 10027254 | | | • | | NT. |
| (II) Meningitis listeria 10027248 Listeria test 10075707 Broad Listeria test positive 10070094 Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Aortitis salmonella 10074937 Arthritis salmonella 10003271 Meningitis salmonella 10027254 | Bacteria | | • | | Narrow |
| Listeria test 10075707 Broad Listeria test positive 10070094 Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Arthritis salmonella 10003271 Meningitis salmonella 10027254 | | | | | _ |
| Listeria test positive 10070094 Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Arthritis salmonella 10003271 Meningitis salmonella 10027254 | | (11) | | | |
| Listeriosis 10024641 Salmonellosis (invasive disease only) (II) Arthritis salmonella 10003271 Meningitis salmonella 10027254 | | | | | Broad |
| Salmonellosis (invasive disease only) (II) Arthritis salmonella Arthritis salmonella Meningitis salmonella 10074937 Narrow Narrow | | | · | | _ |
| disease only) (II) Arthritis salmonella 10003271 Meningitis salmonella 10027254 | | | | | 1 |
| Meningitis salmonella 10027254 | | • | | | Narrow |
| | | disease only) (II) | | | _ |
| Osteomyelitis 10031262 | | | | | _ |
| salmanalla | | | 1 | 10031262 | |
| salmonella Paratyphoid fever 10033971 | | | | 10022071 | $\dashv$ |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Pneumonia salmonella | 10035733 | |
| | | Salmonella bacteraemia | 10058924 | |
| | | Salmonella sepsis | 10058878 | |
| | | Typhoid fever | 10045275 | |
| | | Salmonella test positive | 10070127 | Broad |
| | | Salmonellosis | 10039447 | |
| | | Salmonella test | 10079854 | |
| Bacteria | Shigellosis (invasive | Shigella sepsis | 10074481 | Narrow |
| | disease only) (V) | Shigella infection | 10054178 | Broad |
| | | Shigella test positive | 10070129 | |
| | Vibriosis (invasive | Gastroenteritis vibrio | 10017917 | Broad |
| | disease due to $V$ . | Vibrio test positive | 10070161 | |
| | vulnificus) (V) | None | | Narrow |
| | Infective Pneumonia<br>SMQ | Pneumonia<br>acinetobacter | 10079866 | |
| | | Pneumonia proteus | 10079867 | Narrow |
| | | Pneumonia serratia | 10079868 | |
| Fungal | Aspergillosis (invasive | Aspergillosis oral | 10003489 | |
| | disease only) (II) | Cerebral aspergillosis | 10051597 | |
| | | Meningitis aspergillus | 10073245 | |
| | | Oro-pharyngeal aspergillosis | 10053029 | |
| | | Aspergillus infection | 10074171 | |
| | | Aspergillus test | 10070450 | |
| | | Aspergillus test positive | 10070448 | |
| | | Bronchopulmonary aspergillosis | 10006473 | |
| | | Sinusitis aspergillus | 10051016 | |
| | Blastomycosis (IV) | Blastomycosis | 10005098 | Narrow |
| | | Epididymitis<br>blastomyces | 10015001 | |
| | | Osteomyelitis<br>blastomyces | 10031255 | |
| | | Pneumonia blastomyces | 10035671 | |
| | None | | Broad | |
| | Candidiasis (invasive disease, or oral not | Candida endophthalmitis | 10059449 | Narrow |
| limited to the tongue) (II) | Candida osteomyelitis | 10064699 | | |
| | | Candida pneumonia | 10053158 | |
| | | Candida retinitis | 10068612 | 7 |
| | | Candida sepsis | 10053166 | 7 |
| | | Candida urethritis | 10081262 | 7 |
| | | Candidiasis of trachea | 10064459 | 7 |
| | | Cerebral candidiasis | 10078126 | 7 |
| | | Endocarditis candida | 10014669 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Gastrointestinal candidiasis | 10017938 | |
| | | Hepatic candidiasis | 10049653 | |
| | | Hepatosplenic | 10051590 | 1 |
| | | candidiasis | | |
| | | Meningitis candida | 10027205 | |
| | | Oesophageal candidiasis | 10030154 | |
| | | Oral candidiasis | 10030963 | |
| | | Oropharyngeal candidiasis | 10050346 | |
| | | Peritoneal candidiasis | 10056562 | |
| | | Splenic candidiasis | 10051725 | |
| | | Systemic candida | 10042938 | |
| | | Bladder candidiasis | 10058523 | Broad |
| | | Candida infection | 10074170 | |
| | | Candida test | 10070453 | |
| | | Candida test positive | 10070451 | |
| | | Mucocutaneous candidiasis <sup>1</sup> | 10028080 | |
| | | Respiratory moniliasis | 10038705 | |
| | Coccidioidomycosis (II) | Coccidioides | 10054214 | Narrow |
| | | encephalitis | | |
| | | Coccidioidomycosis | 10009825 | |
| | | Cutaneous coccidioidomycosis | 10068747 | |
| | | Meningitis coccidioides | 10027207 | _ |
| | | None None | 1002/20/ | Broad |
| | Cryptococcosis (II) | Cryptococcal cutaneous infection | 10054216 | Narrow |
| | | Cryptococcal fungaemia | 10067112 | |
| | | Cryptococcosis | 10007112 | _ |
| | | Disseminated | 10013439 | |
| | | cryptococcosis | | |
| | | Gastroenteritis | 10011485 | _ |
| | | cryptococcal Meningitis cryptococcal | 10027209 | |
| | | Neurocryptococcosis | 10027209 | |
| | | Pneumonia cryptococcal | 10067565 | _ |
| | | Cryptococcus test | 10007363 | Broad |
| | | Cryptococcus test Cryptococcus test | 10070436 | |
| | | positive | 100/0433 | |
| | Histoplasmosis (II) | Acute pulmonary | 10001027 | Narrow |
| | | histoplasmosis Chronic pulmonary histoplasmosis | 10009115 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | 22.1) | 10014656 | |
| | | Endocarditis | 10014676 | |
| | | histoplasma | 10020141 | _ |
| | | Histoplasmosis | 10020141 | _ |
| | | Histoplasmosis | 10049142 | |
| | | cutaneous | 10020144 | - |
| | | Histoplasmosis disseminated | 10020144 | |
| | | Meningitis histoplasma | 10027243 | |
| | | Pericarditis histoplasma | 10034489 | |
| | | Retinitis histoplasma | 10038912 | |
| | | Presumed ocular<br>histoplasmosis<br>syndrome | 10063664 | Broad |
| | Microsporidiosis (IV) | Microsporidia infection | 10053982 | Narrow |
| | (* ') | None | | Broad |
| | Other invasive fungi: | Allescheriosis | 10001754 | Narrow |
| | Mucormycosis | Fusarium infection | 10051919 | |
| | (=zygomycosis) | Mucormycosis | 10028098 | |
| | [Rhizopus, Mucor, and | Scedosporium infection | 10059045 | |
| | Lichtheimia], Scedosporum/ | Pseudallescheria infection | 10061919 | |
| | Pseudallescheria boydii, | Pseudallescheria sepsis | 10058973 | |
| | Fusarium (II) | See "Non-specific terms" below | | Broad |
| | Paracoccidioides | Paracoccidioides | 10061906 | Narrow |
| | infections (V) | infection | | |
| | | None | | Broad |
| | Penicillium marneffei | Penicillium infection | 10078580 | Narrow |
| | (V) | None | | Broad |
| | Pneumocystis jirovecii (II) | Pneumocystis jirovecii infection | 10073756 | Narrow |
| | | Pneumocystis jirovecii pneumonia | 10073755 | |
| | | Blood beta-D-glucan | 10068725 | Broad |
| | | Blood beta-D-glucan | 10051795 | |
| | | abnormal | | |
| | | Blood beta-D-glucan | 10051793 | |
| | | increased | | |
| | | Gomori methenamine | 10075549 | |
| | | silver stain | | |
| | | Carbon monoxide | 10065906 | |
| | | diffusing capacity decreased | | |
| | | Carbon monoxide diffusing capacity | 10071738 | |

| test 10070454 |
|------------------------------|
| 10011676 Narrow |
| 10041736 |
| Broad |
| rus 10048843 Narrow |
| rus colitis 10048983 |
| rus 10049014 |
| rus 10049074 |
| rus 10049015 |
| rus 10049016 |
| rus 10051349 |
| rus 10052817 |
| rus 10075619<br>ıl ulcer |
| rus 10011830 |
| rus 10011831 |
| rus 10011834<br>s |
| rus 10065036<br>is ulcer |
| rus 10065621<br>pradiculitis |
| rus 10056261 |
| rus 10079095 |
| rus 10049018 |
| rus 10049566 |
| rus 10056721 |
| rus 10056262 |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Cytomegalovirus<br>urinary tract infection | 10051350 | |
| | | Cytomegalovirus viraemia | 10058854 | |
| | | Disseminated cytomegaloviral infection | 10049075 | |
| | | Encephalitis cytomegalovirus | 10014586 | |
| | | Pneumonia cytomegaloviral | 10035676 | |
| | | Cytomegalovirus test | 10061806 | Broad |
| | | Cytomegalovirus test positive | 10051620 | |
| | HBV reactivation (IV) | None | | Narrow |
| | | Asymptomatic viral hepatitis | 10063838 | Broad |
| | | Chronic hepatitis B | 10008910 | |
| | | HBV-DNA polymerase increased | 10058937 | |
| | | Hepatitis B | 10019731 | |
| | | Hepatitis B antigen | 10063414 | |
| | | Hepatitis B antigen positive | 10063411 | |
| | | Hepatitis B core antigen | 10051160 | |
| | | Hepatitis B core antigen positive | 10052328 | |
| | | Hepatitis B DNA assay | 10060027 | |
| | | Hepatitis B DNA assay positive | 10060047 | |
| | | Hepatitis B DNA increased | 10068379 | |
| | | Hepatitis B e antigen | 10050914 | |
| | | Hepatitis B e antigen positive | 10052329 | |
| | | Hepatitis B reactivation | 10058827 | |
| | | Hepatitis B surface antigen | 10050529 | |
| | | Hepatitis B surface antigen positive | 10019742 | |
| | | Hepatitis B virus test | 10068415 | |
| | | Hepatitis B virus test positive | 10070217 | |
| | | Hepatitis A | 10019780 | |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Hepatitis post transfusion | 10019791 | |
| | | Hepatitis viral | 10019799 | |
| | | Withdrawal hepatitis | 10071220 | |
| Viral | HCV progression (V) | None Withdrawar nepatitis | 100/1220 | Narrow |
| viiai | TIC v progression (v) | Chronic hepatitis C | 10008912 | Broad |
| | | Hepatitis C | 10008912 | Bioau |
| | | • | | _ |
| | | Hepatitis C RNA | 10019748 | _ |
| | | Hepatitis C RNA | 10068727 | |
| | | fluctuation | 100(0277 | _ |
| | | Hepatitis C RNA | 10068377 | |
| | | increased | 10010550 | _ |
| | | Hepatitis C RNA | 10019750 | |
| | | positive | | _ |
| | | Hepatitis C virus test | 10068416 | |
| | | Hepatitis C virus test | 10070218 | |
| | | positive | | |
| | Herpes simplex (IV) | Colitis herpes | 10051782 | Narrow |
| | | Eczema herpeticum | 10014197 | |
| | | Gastritis herpes | 10051784 | |
| | | Herpes oesophagitis | 10052330 | |
| | | Herpes sepsis | 10058876 | |
| | | Herpes simplex colitis | 10074239 | |
| | | Herpes simplex | 10019953 | |
| | | encephalitis | | |
| | | Herpes simplex gastritis | 10074240 | |
| | | Herpes simplex hepatitis | 10067389 | |
| | | Herpes simplex | 10019956 | |
| | | meningitis | | |
| | | Herpes simplex | 10074247 | |
| | | meningoencephalitis | | |
| | | Herpes simplex | 10074250 | |
| | | meningomyelitis | | |
| | | Herpes simplex | 10074252 | |
| | | necrotising retinopathy | | |
| | | Herpes simplex | 10074242 | |
| | oesophagitis | | | |
| | Herpes simplex | 10065046 | | |
| | pneumonia | | | |
| | | Herpes simplex sepsis | 10074246 | |
| | | Herpes simplex visceral | 10019963 | |
| | | Meningitis herpes | 10027242 | |
| | | Meningoencephalitis | 10027285 | |
| | | herpetic | | _ |
| | Meningomyelitis herpes | 10074249 | | |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Pneumonia herpes viral | 10035703 | |
| | | Genital herpes simplex | 10073931 | |
| | | Herpes dermatitis | 10062639 | |
| | | Herpes pharyngitis | 10066888 | |
| | | Herpes simplex otitis externa | 10019959 | |
| | | Herpes simplex pharyngitis | 10074244 | |
| | | Ophthalmic herpes simplex | 10073938 | |
| | | Proctitis herpes | 10036780 | |
| | | Kaposi's varicelliform eruption | 10051891 | |
| | | Herpes simplex test positive | 10077969 | Broad |
| | | Herpes simplex | 10019948 | |
| | | Herpes virus infection | 10019973 | |
| | | Nasal herpes | 10074936 | |
| | | Oral herpes | 10067152 | |
| | | Genital herpes | 10018150 | |
| | Herpes zoster (any form) (II) | Disseminated varicella zoster vaccine virus infection | 10076667 | Narrow |
| | | Encephalitis post varicella | 10014603 | |
| | | Genital herpes zoster | 10072210 | |
| | | Herpes zoster | 10019974 | |
| | | Herpes zoster cutaneous disseminated | 10074297 | |
| | | Herpes zoster disseminated | 10065038 | |
| | | Herpes zoster infection neurological | 10061208 | |
| | | Herpes zoster meningitis | 10074259 | |
| | | Herpes zoster<br>meningoencephalitis | 10074248 | |
| | | Herpes zoster<br>meningomyelitis | 10074251 | |
| | | Herpes zoster<br>meningoradiculitis | 10079327 | |
| | | Herpes zosternecrotising retinopathy | 10074253 | |
| | | Herpes zoster oticus | 10063491 | |
| | | Herpes zoster pharyngitis | 10074245 | |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Necrotising herpetic retinopathy | 10065119 | |
| | | Ophthalmic herpes zoster | 10030865 | |
| | | Varicella | 10046980 | |
| | | Varicella keratitis | 10077496 | |
| | | Varicella post vaccine | 10063522 | |
| | | Varicella zoster gastritis | 10074241 | |
| | | Varicella zoster<br>oesophagitis | 10074243 | |
| | | Varicella zoster pneumonia | 10074254 | |
| | | Varicella zoster virus infection | 10075611 | |
| | | Herpes ophthalmic | 10062004 | |
| | | Varicella virus test | 10070444 | Broad |
| | | Varicella virus test positive | 10070214 | |
| | Human Polyomavirus | BK virus infection | 10055181 | Narrow |
| | infection including BK virus disease and PVAN | Human polyomavirus infection | 10057366 | |
| | (V), and Progressive<br>Multifocal | JC virus granule cell neuronopathy | 10074361 | |
| | Leukoencephalopathy | JC virus infection | 10023163 | |
| | (IV) | Polyomavirus-associated nephropathy | 10065381 | |
| | | Progressive multifocal leukoencephalopathy | 10036807 | |
| | | JC virus test | 10068794 | Broad |
| | | Polyomavirus test | 10075038 | |
| | | Polyomavirus test positive | 10070342 | |
| | Post-transplant<br>lymphoproliferative<br>disorder (EBV) (V) | Epstein-Barr virus<br>associated<br>lymphoproliferative<br>disorder | 10068349 | Narrow |
| | | Post-transplant lymphoproliferative disorder | 10051358 | |
| | | Epstein-Barr viraemia | 10065110 | Broad |
| | | Epstein-Barr virus associated lymphoma | 10071441 | Dioud |
| | | Epstein-Barr virus infection | 10015108 | |

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Lymphoproliferative disorder | 10061232 | |
| | | Lymphoproliferative disorder in remission | 10061233 | |
| | | Oral hairy leukoplakia | 10030979 | |
| Parasites | Trypanosoma cruzi | None | | Narrow |
| | infection (Chagas'<br>Disease) (disseminated | American trypanosomiasis | 10001935 | Broad |
| | disease only) (V) | Trypanosomiasis | 10044707 | |
| | | Meningitis<br>trypanosomal | 10027258 | |
| | Cryptosporidium species (chronic disease only) | Biliary tract infection cryptosporidial | 10067319 | Narrow |
| | (IV) | Cryptosporidiosis infection | 10011502 | Broad |
| | | Gastroenteritis cryptosporidial | 10017899 | |
| | Leishmaniasis (Visceral | Visceral leishmaniasis | 10047505 | Narrow |
| | only) (IV) | Leishmaniasis | 10024198 | Broad |
| (hypsyndiss<br>diss<br>(IV) | Stronglyoides (hyperinfection | None | | Narrow |
| | syndrome and disseminated forms only) | Strongyloidiasis | 10042254 | Broad |
| | Toxoplasmosis (IV) | Cerebral toxoplasmosis | 10057854 | Narrow |
| | | Eye infection toxoplasmal | 10015939 | |
| | | Hepatitis toxoplasmal | 10019798 | |
| | | Meningitis toxoplasmal | 10048848 | |
| | | Myocarditis toxoplasmal | 10028617 | |
| | | Pneumonia toxoplasmal | 10067566 | |
| | | Toxoplasma serology | 10050941 | Broad |
| | | Toxoplasmosis | 10044272 | |
| Non-specific | Non-specific terms | None | | Narrow |
| terms | | Delftia acidovorans | 10081339 | |
| | | Infection | 10081563 | - |
| | | Sphingomonas paucimobilis | 10081303 | |
| | | bacteraemia | | |
| | | Central nervous system immune reconstitution | 10080100 | Broad |
| | | inflammatory response | | |
| | | Abscess fungal | 10000269 | 7 |
| | | Alternaria infection | 10054207 | |
| | | Arthritis fungal | 10060966 | |

| Category | Potential Opportunistic Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| | | Biliary tract infection fungal | 10065203 | |
| | | Central nervous system fungal infection | 10072805 | |
| | | Cerebral fungal infection | 10049657 | |
| | | Encephalitis fungal | 10065170 | |
| | | Erythema induratum | 10015213 | |
| | | Eye infection fungal | 10015933 | |
| | | Fungaemia | 10017523 | |
| | | Fungal abscess central nervous system | 10017524 | |
| | | Fungal endocarditis | 10017529 | |
| | | Fungal labyrinthitis | 10065174 | |
| | | Fungal oesophagitis | 10049656 | |
| | | Fungal peritonitis | 10061138 | |
| | | Fungal pharyngitis | 10076516 | |
| | | Fungal retinitis | 10068613 | |
| | | Fungal sepsis | 10058872 | |
| | | Fungal urethritis | 10081163 | |
| | | Hepatic infection fungal | 10065217 | |
| | | Meningitis fungal | 10027236 | |
| | | Mycotic | 10063202 | |
| | | endophthalmitis | | |
| | | Myocarditis mycotic | 10059026 | |
| | | Oral fungal infection | 10061324 | |
| | | Oropharyngitis fungal | 10061891 | |
| | | Osteomyelitis fungal | 10065239 | |
| | | Otitis media fungal | 10065175 | |
| | | Pancreatitis fungal | 10065190 | |
| | | Pericarditis fungal | 10065220 | |
| | | Phaehyphomycosis | 10034799 | |
| | | Pneumonia fungal | 10061354 | |
| | | Pulmonary mycosis | 10037422 | |
| | | Pulmonary | 10068184 | |
| | | trichosporonosis | | |
| | | Sinusitis fungal | 10058678 | |
| | | Splenic infection fungal | 10065194 | |
| | | Systemic mycosis | 10052366 | |
| | Infective Pneumonia | All PTs (exclude | | |
| Pneumonia | | COVID-19 and | 20000231 | Narrow |
| | SMQ | influenza PTs) | | |

Abbreviations: DNA = deoxyribonucleic acid; EBV= Epstein-Barr virus; HBV = hepatitis B virus; MedDRA = Medical Dictionary for Regulatory Activities; PT = Preferred Term; PVAN = Polyomavirus-associated nephropathy; SMQ = Standardized MedDRA Query.

# Appendix 5. List of MedDRA Preferred Terms for Elevated or Increased Lipids from the Dyslipidemia SMQ (SMQ 20000026)

| Preferred Term (MedDRA Version 20.0) | Preferred Term Code |
|-----------------------------------------------------|---------------------|
| Apolipoprotein B/Apolipoprotein A-1 ratio increased | 10065516 |
| Autoimmune hyperlipidaemia | 10071577 |
| Blood cholesterol abnormal | 10005423 |
| Blood cholesterol increased | 10005425 |
| Blood triglycerides abnormal | 10005837 |
| Blood triglycerides increased | 10005839 |
| Diabetic dyslipidaemia | 10070901 |
| Dyslipidaemia | 10058108 |
| Familial hypertriglyceridaemia | 10059183 |
| Fat overload syndrome | 10074028 |
| High density lipoprotein abnormal | 10020051 |
| High density lipoprotein decreased | 10020060 |
| High density lipoprotein increased | 10020061 |
| Hypercholesterolaemia | 10020603 |
| Hyperlipidaemia | 10062060 |
| Hypertriglyceridaemia | 10020869 |
| Hypo HDL cholesterolaemia | 10068961 |
| Intermediate density lipoprotein increased | 10064236 |
| LDL/HDL ratio increased | 10049030 |
| Lipid metabolism disorder | 10061227 |
| Lipids abnormal | 10024588 |
| Lipids increased | 10024592 |
| Lipoprotein (a) abnormal | 10054023 |
| Lipoprotein (a) increased | 10054009 |
| Low density lipoprotein abnormal | 10024901 |
| Low density lipoprotein increased | 10024910 |
| Non-high-density lipoprotein cholesterol increased | 10063967 |
| Remnant hyperlipidaemia | 10038316 |
| Total cholesterol/HDL ratio abnormal | 10058633 |
| Total cholesterol/HDL ratio increased | 10058630 |

| Preferred Term (MedDRA Version 20.0) | Preferred Term Code |
|----------------------------------------|---------------------|
| Type I hyperlipidaemia | 10060749 |
| Type II hyperlipidaemia | 10045254 |
| Type IIa hyperlipidaemia | 10045261 |
| Type IIb hyperlipidaemia | 10045263 |
| Type III hyperlipidaemia | 10060751 |
| Type IV hyperlipidaemia | 10060753 |
| Type V hyperlipidaemia | 10060755 |
| Very low density lipoprotein abnormal | 10047352 |
| Very low density lipoprotein increased | 10047361 |

Abbreviation: MedDRA = Medical Dictionary for Regulatory Activities.

## Appendix 6. List of Planned Laboratory Analytes with Reference Range Sources

| Laboratory | Laboratory Analyte | Reference | Analysis Type | |
|---|---|---|---|---|
| Group/Order | | Range Name | Central | Outlier/Shift |
| | | | Tendency | Analysis |
| Hematology | | | | |
| 1 | Hemoglobin | LCTPB | Yes | Yes |
| 2 | Hematocrit | LCTPB | Yes | Yes |
| 3 | Erythrocyte Count | LCTPB | Yes | Yes |
| 4 | Mean Cell Volume | LCTPB | Yes | Yes |
| 5 | Mean Cell Hemoglobin | LCTPB | Yes | Yes |
| 6 | MCHC | LCTPB | Yes | Yes |
| 7 | Platelets | LCTPB | Yes | Yes |
| 8 | Leukocyte Count | LCTPB | Yes | Yes |
| 9 | Bands | LCTPB | Yes | Yes |
| 10 | Neutrophils | LCTPB | Yes | Yes |
| 11 | Lymphocytes | LCTPB | Yes | Yes |
| 12 | Monocytes | LCTPB | Yes | Yes |
| 13 | Eosinophils | LCTPB | Yes | Yes |
| 14 | Basophils | LCTPB | Yes | Yes |
| Chemistry | | | | |
| 1 | ALT/SGPT | Covance | Yes | Yes |
| 2 | AST/SGOT | Covance | Yes | Yes |
| 3 | Alkaline Phosphatase | Covance | Yes | Yes |
| 4 | Total Bilirubin | Covance | Yes | Yes |
| 5 | Direct Bilirubin | Covance | Yes | Yes |
| 6 | Albumin | LCTPB | Yes | Yes |
| 7 | Creatine Phosphokinase | LCTPB | Yes | Yes |
| 8 | Creatinine | Covance | Yes | Yes |
| 9 | Urea Nitrogen | LCTPB | Yes | Yes |
| 11 | estimated GFR | Covance | Yes | Yes |
| 12 | Creatinine Clearance | Covance | Yes | Yes |
| 13 | Sodium | LCTPB | Yes | Yes |
| 14 | Potassium | LCTPB | Yes | Yes |
| 15 | Calcium | LCTPB | Yes | Yes |
| 16 | Total Protein | LCTPB | Yes | Yes |
| 17 | Fasting Glucose | LCTPB | Yes | Yes |
| 18 | Glucose, Non-Fasting or Random | LCTPB | Yes | Yes |
| 19 | Uric Acid | LCTPB | Yes | Yes |
| 20 | Cholesterol | LCTPB | Yes | Yes |
| 21 | Triglycerides | LCTPB | Yes | Yes |
| 22 | LDL Cholesterol – Direct | Covance | Yes | Yes |
| 23 | HDL Cholesterol – Direct | Covance | Yes | Yes |
| 24 | LDL/HDL Ratio – Calculated | None | Yes | No |

| Laboratory | Laboratory Analyte | Reference | Analysis Type | |
|---|---|---|---|---|
| Group/Order | | Range Name | Central<br>Tendency | Outlier/Shift<br>Analysis |
| Immunoglobu | lins | | | |
| 1 | Immunoglobulin A | Covance | Yes | Yes |
| 2 | Immunoglobulin G | Covance | Yes | Yes |
| 3 | Immunoglobulin M | Covance | Yes | Yes |
| Urinalysis | | | | |
| 1 | Specific Gravity | LCTPB | Yes | Yes |
| 2 | pН | LCTPB | Yes | Yes |
| 3 | UA-color | None | No | Yes |
| 4 | UA-glucose | None | No | Yes |
| 5 | UA-protein | None | No | Yes |
| 6 | UA-bilirubin | None | No | Yes |
| 7 | UA-urobilinogen | None | No | Yes |
| 8 | UA-nitrites | None | No | Yes |
| 9 | UA-leukoesterase | None | No | Yes |
| 10 | UA-ketones | None | No | Yes |
| 11 | UA-occult blood | None | No | Yes |





Abbreviations: ALT/SGPT = alanine aminotransferase/serum glutamic pyruvic transaminase;

AST/SGOT = aspartate aminotransferase/serum glutamic oxaloacetic transaminase; CD = cluster of differentiation; HDL = high-density lipoprotein; Ig = immunoglobulin; LCTPB = Lilly Large Clinical Trial Population Based; LDL = low-density lipoprotein; MCHC = mean corpuscular hemoglobin concentration;

UA = urinalysis.

#### **Appendix 7. Common Terminology Criteria for Adverse Events (CTCAE) Related to Myelosuppressive Events**

| | Laboratory | | | |
|---|---|---|---|---|
| Event | Test | Grade | Criteria in Système International (SI) Units | Criteria in Conventional (CN) Units |
| Anemia <sup>a</sup> | Hemoglobin | 0 (normal) | ≥7.27 mmol (Fe)/L for females and ≥8.18 mmol (Fe)/L for males | ≥12 g/dL for females and ≥13.5 g/dL for males |
| | | 1 | <7.27 mmol (Fe)/L for females and 8.18 mmol (Fe)/L for males and ≥6.2 mmol (Fe)/L | <12 g/dL for females and 13.5 g/dL for males and $\geq$ 10 g/dL |
| | | 2 | $<$ 6.2 mmol (Fe)/L and $\ge$ 4.9 mmol (Fe)/L | $<10 \text{ g/dL}$ and $\ge 8.0 \text{ g/dL}$ |
| | | 3 | <4.9 mmol (Fe)/L and ≥4.0 mmol (Fe)/L | $<$ 8.0 g/dL and $\ge$ 6.5 g/dL |
| | | 4 | <4.0 mmol (Fe)/L | <6.5 g/dL |
| Leukopenia <sup>a</sup> | White blood | 0 (normal) | ≥4.0 billion cells/L | ≥4.0 thousand cells/uL |
| | cell (WBC) | 1 | <4.0 billion cells/L and ≥3.0 billion cells/L | <4.0 thousand cells/uL and ≥3.0 thousand cells/uL |
| | count | 2 | <3.0 billion cells/L and ≥2.0 billion cells/L | <3.0 thousand cells/uL and ≥2.0 thousand cells/uL |
| | | 3 | $<$ 2.0 billion cells/L and $\ge$ 1.0 billion cells/L | <2.0 thousand cells/uL and ≥1.0 thousand cells/uL |
| | | 4 | <1.0 billion cells/L | <1.0 thousand cells/uL |
| Neutropeniaa | Absolute | 0 (normal) | ≥2 billion cells/L | ≥2 thousand cells/uL |
| | neutrophil | 1 | <2 billion cells/L and ≥1.5 billion cells/L | <2 thousand cells/uL and ≥1.5 thousand cells/uL |
| | count (ANC) | 2 | <1.5 billion cells/L and ≥1.0 billion cells/L | $<$ 1.5 thousand cells/uL and $\ge$ 1.0 thousand cells/uL |
| | | 3 | $<$ 1.0 billion cells/L and $\ge$ 0.5 billion cells/L | <1.0 thousand cells/uL and ≥0.5 thousand cells/uL |
| | | 4 | <0.5 billion cells/L | <0.5 thousand cells/uL |
| Lymphopeniaa | Lymphocyte | 0 (normal) | ≥1.1 billion cells/L | ≥1.1 thousand cells/uL |
| | count | 1 | <1.1 billion cells/L and ≥0.8 billion cells/L | <1.1 thousand cells/uL and ≥0.8 thousand cells/uL |
| | | 2 | $<$ 0.8 billion cells/L and $\ge$ 0.5 billion cells/L | <0.8 thousand cells/uL and ≥0.5 thousand cells/uL |
| | | 3 | $<$ 0.5 billion cells/L and $\ge$ 0.2 billion cells/L | $<$ 0.5 thousand cells/uL and $\ge$ 0.2 thousand cells/uL |
| | | 4 | <0.2 billion cells/L | <0.2 thousand cells/uL |
| Thrombocytopeniaa | Platelet count | 0 (normal) | ≥150 billions/L | ≥150 thousands/uL |
| | | 1 | <150 billions/L and ≥75 billions/L | <150 thousands/uL and ≥75 thousands/uL |
| | | 2 | <75 billions/L and ≥50 billions/L | <75 thousands/uL and ≥50 thousands/uL |
| | | 3 | <50 billions/L and ≥25 billions/L | <50 thousands/uL and ≥25 thousands/uL |
| | | 4 | <25 billions/L | <25 thousands/uL |

Abbreviation: CTCAE = Common Terminology Criteria for Adverse Events; Fe = iron.

a CTCAE grading was adjusted by replacing lower limit of normal (LLN) with a single value.

#### Signature Page for VV-CLIN-074563 v1.0

| Approval | PPD |
|----------|-------------------------------|
| | 31-Jan-2023 18:28:13 GMT+0000 |

Signature Page for VV-CLIN-074563 v1.0